CLINICAL TRIAL: NCT00676403
Title: Randomized, Double-Blind, 6-Week Study Of Pregabalin In Subjects With Restless Legs Syndrome
Brief Title: Lyrica Dose Response Study With Restless Legs Syndrome (RLS) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081183
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2010-06

CONDITIONS: Restless Legs Syndrome
Keywords: pregabalin, RLS, efficacy, safety
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Sugars; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- 2 (Experimental): investigational treatment
  Interventions: Drug: Pregabalin
- 3 (Experimental): investigational treatment
  Interventions: Drug: Pregabalin
- 4 (Experimental): investigational treatment
  Interventions: Drug: Pregabalin
- 5 (Experimental): investigational treatment
  Interventions: Drug: Pregabalin
- 6 (Experimental): investigational treatment
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: placebo — Placebo control (capsule), once a day, 1- 3 hours before bedtime for 6 weeks
  Other Names: Sugar pill
  Arms: 1
Drug: Pregabalin — 50 mg (capsule) per day, 1 - 3 hours before bedtime for 6 weeks
  Other Names: Lyrica, PD 0144723; CI-1008
  Arms: 2
Drug: Pregabalin — 100 mg (capsule) per day, 1 - 3 hours before bedtime for 6 weeks
  Other Names: Lyrica, PD 0144723; CI-1008
  Arms: 3
Drug: Pregabalin — 150 mg (capsule) per day, 1 - 3 hours before bedtime for 6 weeks
  Other Names: Lyrica, PD 0144723; CI-1008
  Arms: 4
Drug: Pregabalin — 300 mg (capsule) per day, 1 - 3 hours before bedtime for 6 weeks
  Other Names: Lyrica, PD 0144723; CI-1008
  Arms: 5
Drug: Pregabalin — 450 mg (capsule) per day, 1 - 3 hours before bedtime for 6 weeks
  Other Names: Lyrica, PD 0144723; CI-1008
  Arms: 6

SUMMARY:
To test the effectiveness and tolerability of Lyrica at various dose levels in RLS patients

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe idiopathic RLS
* symptoms occur predominantly in the evening
* symptoms interfere with sleep onset or maintenance

Exclusion Criteria:

* Any secondary RLS
* require treatment for daytime RLS symptoms
* symptomatic neuropathies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (15):
  - Pfizer Investigational Site, Tuscaloosa, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Brandon, Florida
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Alexandria, Virginia
- Austria (2):
  - Pfizer Investigational Site, Innsbruck
  - Pfizer Investigational Site, Vienna
- Germany (7):
  - Pfizer Investigational Site, Bad Saarow
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Mittweida
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Oldenburg
  - Pfizer Investigational Site, Schwerin
- Pfizer Investigational Site, Madrid, Spain

REFERENCES:
- [Derived] Allen R, Chen C, Soaita A, Wohlberg C, Knapp L, Peterson BT, Garcia-Borreguero D, Miceli J. A randomized, double-blind, 6-week, dose-ranging study of pregabalin in patients with restless legs syndrome. Sleep Med. 2010 Jun;11(6):512-9. doi: 10.1016/j.sleep.2010.03.003. Epub 2010 May 13. PMID 20466589
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081183&StudyName=Lyrica%20Dose%20Response%20Study%20With%20Restless%20Legs%20Syndrome%20%28RLS%29%20patients

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects meeting entry criteria with a confirmed diagnosis of Restless Leg Syndrome completed a washout of medications if needed prior to starting a 7-day single-blind placebo run-in to identify and exclude placebo responders and to adapt subjects to take study drug 1-3 hours prior to bedtime. Of 218 subjects screened, 137 subjects entered.
Groups:
- Placebo: Single daily oral dose.
- Pregabalin 50 mg: Single daily 50 mg oral dose.
- Pregabalin 100 mg: Single daily 100 mg oral dose. Dose was escalated from 50 mg/day after Day 3.
- Pregabalin 150 mg: Single daily 150 mg oral dose. Dose was escalated from 75 mg/day after Day 3.
- Pregabalin 300 mg: Single daily 300 mg oral dose. Dose was escalated from 75 mg/day (Days 1-3), and 150 mg/day (Days 4-7).
- Pregabalin 450 mg: Single daily 450 mg oral dose. Dose was escalated from 75 mg/day (Days 1-3), 150 mg/day (Days 4-7), and 300 mg/day (Days 8-11).
Period: Overall Study
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Started | 23 | 22 | 23 | 22 | 24 | 23
Completed | 21 | 20 | 22 | 17 | 23 | 18
Not Completed | 2 | 2 | 1 | 5 | 1 | 5
Not completed — Adverse Event | 1 | 2 | 0 | 5 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Reason Unspecified | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg | Total
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23 | 137
Age, Customized [Number; unit: participants]
  18 - 44 years | 4 | 5 | 7 | 2 | 9 | 3 | 30
  45 - 64 years | 19 | 15 | 16 | 20 | 15 | 19 | 104
  >=65 years | 0 | 2 | 0 | 0 | 0 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 16 | 13 | 19 | 16 | 90
  Male | 10 | 9 | 7 | 9 | 5 | 7 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Restless Leg Syndrome (RLS) International Restless Leg Group Symptom Severity Rating Scale (IRLS) Total Score at Week 6
Description: IRLS: Subject-rated instrument to assess RLS symptom severity and impact on daily living; 10 items yielding 2 subscale scores and 1 global (total) score. Subscale scores: symptom severity (6 items) and impact on daily living (3 items), with item 5 (daytime somnolence due to RLS) loaded equally on both subscales. Global score: calculated from all 10 items. Subscale score ranges: symptom severity 0-24, impact of daily living 0-12; global score range: 0-40. Lower scores reflect lower severity and better quality of life. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 6
Population: ITT. Baseline statistics were calculated only for subjects who had a non-missing change from baseline at at least one post-baseline visit. Recall period = week prior to assessment.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 21 | 20 | 22 | 18 | 23 | 20
scores on scale | -7.73 (1.720) | -11.83 (1.771) | -11.76 (1.694) | -16.02 (1.865) | -12.89 (1.713) | -16.26 (1.771)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg vs Pregabalin 100 mg vs Pregabalin 150 mg vs Pregabalin 300 mg vs Pregabalin 450 mg; Dose response analysis ED 50: dose providing 50% of the maximal effect. Statistics were obtained from three parameter model Y = D + G*exp(B*dose) by bootstrapping 2000 data sets, where D = expected response of saturation (maximal effect), B = related to slope of the dose response mechanism (change in response relative to the change in dose), and D+G = expected response at zero dose; Test type: Superiority or Other; ED-50: Bootstrap Method; Median Difference (Final Values) = 37.3, 95% CI [0.1 to 157.7] — Non-convergence for the non-liner model occurred in some bootstrap samples which were not included in summarizing the ED50 distribution or confidence interval
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 50 mg vs Pregabalin 100 mg vs Pregabalin 150 mg vs Pregabalin 300 mg vs Pregabalin 450 mg; Dose response analysis ED 90: dose providing 90% of the maximal effect. Statistics were obtained from three parameter model Y = D + G*exp(B*dose) by bootstrapping 2000 data sets, where D = expected response of saturation (maximal effect), B = related to slope of the dose response mechanism (change in response relative to the change in dose), and D+G = expected response at zero dose; Test type: Superiority or Other; ED 90: Bootstrap Method; Median Difference (Final Values) = 123.9, 95% CI [0.4 to 523.9] — Non-convergence for the non-liner model occurred in some bootstrap samples which were not included in summarizing the ED90 distribution or confidence interval
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 50 mg; Week 6: Contrast of treatment vs. placebo. The repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score was included as a covariate. Additionally, model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.0983, Mixed Models Analysis; Mean Difference (Final Values) = -4.10, 95% CI [-8.97 to 0.77], Standard Error of Mean 2.472
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0966, Mixed Models Analysis; Mean Difference (Final Values) = -4.03, 95% CI [-8.78 to 0.73], Standard Error of Mean 2.415
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; Mean Difference (Final Values) = -8.29, 95% CI [-13.31 to -3.28], Standard Error of Mean 2.548
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0353, Mixed Models Analysis; Mean Difference (Final Values) = -5.16, 95% CI [-9.96 to -0.36], Standard Error of Mean 2.437
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Final Values) = -8.53, 95% CI [-13.40 to -3.67], Standard Error of Mean 2.469

2. Secondary Outcome: Number of Subjects Responding to Treatment as Assessed by the Clinical Global Impression - Improvement Scale (CGI-I)
Description: Clinical Global Impression - Improvement Scale (CGI-I): 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected. Number of subjects responding to treatment at Week 6 with respect to dose level. CGI-I Responders = subjects who reported CGI-I scores of very much improved or much improved.
Time Frame: Week 6
Population: ITT; N=number of subjects in a treatment group; n=number of subjects with a clinical Global Impressions Improvement (CGI-I) rating.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
participants
  Week 6: Responders (n=21, 20, 22, 18, 23, 20) | 13 | 12 | 15 | 11 | 17 | 18
  Week 6: Non-Responders | 8 | 8 | 7 | 7 | 6 | 2
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; Week 6: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.8784, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; Week 6: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.6767, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; Week 6: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.8955, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; Week 6: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.9505, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; Week 6: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.0466, Cochran-Mantel-Haenszel

3. Secondary Outcome: Number of Subjects With Categorical Scores on the Clinical Global Impression - Severity Scale (CGI-S)
Description: CGI-S Scale: 7-point clinician rated scale to assess severity of subject's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6, Last Observation Carried Forward (LOCF)
Population: ITT; N=number of subjects in a treatment group. LOCF: Last Observation Carried Forward.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
participants
  Baseline: Normal, Not at All Ill | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: Borderline, Mentally Ill | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: Mildly Ill | 1 | 1 | 2 | 4 | 2 | 2
  Baseline: Moderately Ill | 6 | 9 | 8 | 5 | 11 | 6
  Baseline: Markedly Ill | 7 | 8 | 7 | 5 | 3 | 5
  Baseline: Severely Ill | 8 | 3 | 6 | 7 | 8 | 10
  Baseline: Among the Most Extremely Ill | 1 | 1 | 0 | 1 | 0 | 0
  Week 1: Normal, Not at All Ill | 1 | 1 | 1 | 1 | 0 | 3
  Week 1: Borderline, Mentally Ill | 0 | 1 | 1 | 1 | 4 | 2
  Week 1: Mildly Ill | 4 | 6 | 5 | 8 | 5 | 7
  Week 1: Moderately Ill | 10 | 8 | 5 | 7 | 6 | 8
  Week 1: Markedly Ill | 4 | 3 | 5 | 1 | 3 | 2
  Week 1: Severely Ill | 4 | 2 | 3 | 2 | 5 | 1
  Week 1: Among the Most Extremely Ill | 0 | 0 | 0 | 0 | 0 | 0
  Week 2: Normal, Not at All Ill | 0 | 2 | 1 | 2 | 3 | 7
  Week 2: Borderline, Mentally Ill | 3 | 4 | 2 | 3 | 6 | 2
  Week 2: Mildly Ill | 10 | 5 | 9 | 7 | 4 | 8
  Week 2: Moderately Ill | 3 | 5 | 5 | 6 | 5 | 3
  Week 2: Markedly Ill | 3 | 3 | 4 | 0 | 3 | 0
  Week 2: Severely Ill | 3 | 1 | 1 | 1 | 1 | 0
  Week 2: Among the Most Extremely Ill | 1 | 0 | 0 | 0 | 0 | 0
  Week 4: Normal, Not at All Ill | 1 | 2 | 2 | 5 | 4 | 8
  Week 4: Borderline, Mentally Ill | 4 | 2 | 2 | 2 | 6 | 5
  Week 4: Mildly Ill | 8 | 7 | 11 | 5 | 4 | 4
  Week 4: Moderately Ill | 4 | 6 | 6 | 5 | 5 | 2
  Week 4: Markedly Ill | 3 | 2 | 1 | 1 | 2 | 1
  Week 4: Severely Ill | 2 | 2 | 1 | 1 | 2 | 0
  Week 4: Among the Most Extremely Ill | 0 | 0 | 0 | 0 | 0 | 0
  Week 6: Normal, Not at All Ill | 1 | 3 | 4 | 4 | 6 | 7
  Week 6: Borderline, Mentally Ill | 3 | 3 | 4 | 4 | 4 | 5
  Week 6: Mildly Ill | 11 | 6 | 7 | 7 | 7 | 6
  Week 6: Moderately Ill | 2 | 5 | 5 | 3 | 1 | 1
  Week 6: Markedly Ill | 2 | 2 | 2 | 0 | 4 | 1
  Week 6: Severely Ill | 2 | 1 | 0 | 0 | 1 | 0
  Week 6: Among the Most Extremely Ill | 0 | 0 | 0 | 0 | 0 | 0
  LOCF: Normal | 1 | 3 | 4 | 4 | 6 | 7
  LOCF: Borderline, Mentally Ill | 3 | 3 | 4 | 4 | 4 | 6
  LOCF: Mildly Ill | 12 | 6 | 7 | 9 | 7 | 7
  LOCF: Moderately Ill | 2 | 6 | 5 | 5 | 1 | 1
  LOCF: Markedly Ill | 2 | 2 | 2 | 0 | 4 | 1
  LOCF: Severely Ill | 2 | 2 | 1 | 0 | 2 | 1
  LOCF: Among the Most Extremely Ill | 1 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; Week 1: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.3876, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; Week 1: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.7959, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; Week 1: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.2032, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; Week 1: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.7032, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; Week 1: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.0551, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; Week 2: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.4100, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; Week 2: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.6524, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; Week 2: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.3219, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; Week 2: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.3509, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; Week 2: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.0053, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; Week 4: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.9835, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; Week 4: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.6668, Cochran-Mantel-Haenszel
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; Week 4: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.2823, Cochran-Mantel-Haenszel
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; Week 4: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.5687, Cochran-Mantel-Haenszel
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; Week 4: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.0043, Cochran-Mantel-Haenszel
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; Week 6: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.8662, Cochran-Mantel-Haenszel
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; Week 6: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.3656, Cochran-Mantel-Haenszel
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; Week 6: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.0806, Cochran-Mantel-Haenszel
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; Week 6: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.5381, Cochran-Mantel-Haenszel
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; Week 6: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.0090, Cochran-Mantel-Haenszel
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 50 mg; Last Observation Carried Forward: Cochran-Mantel-Haenszel test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.9748, Cochran-Mantel-Haenszel
Statistical Analysis 22: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.3936, Cochran-Mantel-Haenszel
Statistical Analysis 23: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.1563, Cochran-Mantel-Haenszel
Statistical Analysis 24: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.6357, Cochran-Mantel-Haenszel
Statistical Analysis 25: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.0133, Cochran-Mantel-Haenszel

4. Secondary Outcome: Subjective Sleep Questionnaire (SSQ): Latency Subscale; Observed Change From Baseline
Description: Subjective Sleep Questionnaire (SSQ): subject-rated instrument used to assess sleep behavior; measures sleep quantity and quality. Comprised of 5 items yielding 5 subscale scores: latency, hours of sleep, number of awakenings, total wake time after sleep onset, and quality of sleep. Latency subscale (time to fall asleep [in minutes]): numerical rating completed by the subject 30 minutes after waking; recall period is the night before. Lower score reflects greater ease (shorter time) in falling asleep. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
Population: ITT; baseline statistics were calculated only for subjects who had non-missing change from baseline at at least one post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
minutes
  Week 1 | -9.8 (5.60) | -16.3 (5.76) | -13.2 (5.60) | -10.4 (5.76) | -9.1 (5.65) | -20.2 (5.62)
  Week 2 | -8.9 (5.60) | -20.7 (5.84) | -17.2 (5.65) | -16.3 (6.00) | -13.0 (5.71) | -34.3 (5.69)
  Week 3 | -14.6 (5.71) | -18.9 (5.90) | -13.1 (5.60) | -17.8 (6.00) | -17.8 (5.71) | -33.7 (5.88)
  Week 4 | -13.6 (5.66) | -20.4 (5.90) | -20.4 (5.60) | -18.2 (6.00) | -18.2 (5.71) | -37.1 (5.82)
  Week 5 | -15.9 (5.71) | -26.8 (5.90) | -17.6 (5.60) | -24.0 (6.07) | -13.4 (5.71) | -36.1 (5.82)
  Week 6 | -12.4 (5.71) | -25.4 (5.90) | -19.5 (5.65) | -25.1 (6.14) | -10.1 (5.71) | -34.9 (5.82)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; Week 1: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score was included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.4133, Mixed Models Analysis; Mean Difference (Final Values) = -6.6, 95% CI [-22.4 to 9.3], Standard Error of Mean 8.05
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; Week 1: Conrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score was included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.6676, Mixed Models Analysis; Mean Difference (Final Values) = -3.4, 95% CI [-19.0 to 12.2], Standard Error of Mean 7.92
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9355, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI [-16.5 to 15.2], Standard Error of Mean 8.04
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9355, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI [-15.1 to 16.4], Standard Error of Mean 7.97
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1895, Mixed Models Analysis; Mean Difference (Final Values) = -10.5, 95% CI [-26.1 to 5.2], Standard Error of Mean 7.94
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; Week 2: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score was included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.1443, Mixed Models Analysis; Mean Difference (Final Values) = -11.9, 95% CI [-27.8 to 4.1], Standard Error of Mean 8.10
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.2946, Mixed Models Analysis; Mean Difference (Final Values) = -8.4, 95% CI [-24.0 to 7.3], Standard Error of Mean 7.96
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.3686, Mixed Models Analysis; Mean Difference (Final Values) = -7.4, 95% CI [-23.6 to 8.8], Standard Error of Mean 8.22
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.6079, Mixed Models Analysis; Mean Difference (Final Values) = -4.1, 95% CI [-19.9 to 11.7], Standard Error of Mean 8.02
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 6]; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; Mean Difference (Final Values) = -25.5, 95% CI [-41.2 to -9.7], Standard Error of Mean 7.99
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; Week 3: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score was included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.5976, Mixed Models Analysis; Mean Difference (Final Values) = -4.3, 95% CI [-20.5 to 11.8], Standard Error of Mean 8.22
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.8527, Mixed Models Analysis; Mean Difference (Final Values) = 1.5, 95% CI [-14.3 to 17.3], Standard Error of Mean 8.00
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.6973, Mixed Models Analysis; Mean Difference (Final Values) = -3.2, 95% CI [-19.6 to 13.1], Standard Error of Mean 8.29
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.6895, Mixed Models Analysis; Mean Difference (Final Values) = -3.2, 95% CI [-19.2 to 12.7], Standard Error of Mean 8.09
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 11]; Test type: Superiority or Other; p = 0.0209, Mixed Models Analysis; Mean Difference (Final Values) = -19.1, 95% CI [-35.2 to -2.9], Standard Error of Mean 8.21
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; Week 4: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score was included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.4084, Mixed Models Analysis; Mean Difference (Final Values) = -6.8, 95% CI [-22.9 to 9.3], Standard Error of Mean 8.18
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.3958, Mixed Models Analysis; Mean Difference (Final Values) = -6.8, 95% CI [-22.5 to 8.9], Standard Error of Mean 7.96
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.5776, Mixed Models Analysis; Mean Difference (Final Values) = -4.6, 95% CI [-20.9 to 11.7], Standard Error of Mean 8.25
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.5665, Mixed Models Analysis; Mean Difference (Final Values) = -4.6, 95% CI [-20.5 to 11.3], Standard Error of Mean 8.06
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis; Mean Difference (Final Values) = -23.5, 95% CI [-39.6 to -7.5], Standard Error of Mean 8.13
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 50 mg; Week 5: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score was included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.1842, Mixed Models Analysis; Mean Difference (Final Values) = -10.9, 95% CI [-27.1 to 5.2], Standard Error of Mean 8.22
Statistical Analysis 22: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 4, analysis 21]; Test type: Superiority or Other; p = 0.8269, Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI [-17.5 to 14.0], Standard Error of Mean 8.00
Statistical Analysis 23: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 4, analysis 21]; Test type: Superiority or Other; p = 0.3319, Mixed Models Analysis; Mean Difference (Final Values) = -8.1, 95% CI [-24.5 to 8.3], Standard Error of Mean 8.34
Statistical Analysis 24: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 21]; Test type: Superiority or Other; p = 0.7552, Mixed Models Analysis; Mean Difference (Final Values) = 2.5, 95% CI [-13.4 to 18.5], Standard Error of Mean 8.09
Statistical Analysis 25: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 21]; Test type: Superiority or Other; p = 0.0137, Mixed Models Analysis; Mean Difference (Final Values) = -20.3, 95% CI [-36.3 to -4.2], Standard Error of Mean 8.16
Statistical Analysis 26: Comparison: Placebo vs Pregabalin 50 mg; Week 6: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score was included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.1157, Mixed Models Analysis; Mean Difference (Final Values) = -13.0, 95% CI [-29.2 to 3.2], Standard Error of Mean 8.22
Statistical Analysis 27: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 4, analysis 26]; Test type: Superiority or Other; p = 0.3791, Mixed Models Analysis; Mean Difference (Final Values) = -7.1, 95% CI [-22.9 to 8.7], Standard Error of Mean 8.04
Statistical Analysis 28: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 4, analysis 26]; Test type: Superiority or Other; p = 0.1329, Mixed Models Analysis; Mean Difference (Final Values) = -12.7, 95% CI [-29.2 to 3.9], Standard Error of Mean 8.39
Statistical Analysis 29: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 4, analysis 26]; Test type: Superiority or Other; p = 0.7723, Mixed Models Analysis; Mean Difference (Final Values) = 2.3, 95% CI [-13.6 to 18.3], Standard Error of Mean 8.09
Statistical Analysis 30: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 4, analysis 26]; Test type: Superiority or Other; p = 0.0063, Mixed Models Analysis; Mean Difference (Final Values) = -22.5, 95% CI [-38.6 to -6.4], Standard Error of Mean 8.16

5. Secondary Outcome: Subjective Sleep Questionnaire: Hours of Sleep Subscale; Observed Change From Baseline
Description: Subjective Sleep Questionnaire (SSQ): subject-rated instrument used to assess sleep behavior; measures sleep quantity and quality. Comprised of 5 items yielding 5 subscale scores: latency, hours of sleep, number of awakenings, total wake time after sleep onset, and quality of sleep. Hours of sleep subscale reflects change in hours of sleep from baseline. Numerical rating completed by the subject 30 minutes after waking; recall period is the night before.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
Population: ITT; baseline statistics were calculated only for subjects who had a non-missing change from baseline at at least one post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
hours
  Week 1 | 0.23 (0.177) | 0.57 (0.183) | 0.29 (0.177) | 0.55 (0.182) | 0.45 (0.177) | 0.72 (0.178)
  Week 2 | 0.36 (0.177) | 0.65 (0.186) | 0.52 (0.179) | 0.81 (0.192) | 0.76 (0.180) | 1.07 (0.181)
  Week 3 | 0.36 (0.182) | 0.61 (0.188) | 0.53 (0.177) | 0.89 (0.192) | 0.72 (0.180) | 1.32 (0.189)
  Week 4 | 0.27 (0.180) | 0.81 (0.188) | 0.46 (0.177) | 0.93 (0.192) | 0.65 (0.180) | 1.03 (0.187)
  Week 5 | 0.37 (0.182) | 1.03 (0.188) | 0.43 (0.177) | 0.97 (0.195) | 0.61 (0.180) | 1.43 (0.187)
  Week 6 | 0.19 (0.182) | 0.84 (0.188) | 0.42 (0.179) | 0.95 (0.198) | 0.44 (0.180) | 1.11 (0.187)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; Week 1: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score is included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.1715, Mixed Models Analysis; Mean Difference (Final Values) = 0.35, 95% CI [-0.15 to 0.85], Standard Error of Mean 0.254
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.7944, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI [-0.43 to 0.56], Standard Error of Mean 0.251
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1994, Mixed Models Analysis; Mean Difference (Final Values) = 0.33, 95% CI [-0.17 to 0.83], Standard Error of Mean 0.255
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.3652, Mixed Models Analysis; Mean Difference (Final Values) = 0.23, 95% CI [-0.27 to 0.72], Standard Error of Mean 0.251
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0481, Mixed Models Analysis; Mean Difference (Final Values) = 0.50, 95% CI [0.00 to 0.99], Standard Error of Mean 0.251
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; Week 2: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score is included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.2501, Mixed Models Analysis; Mean Difference (Final Values) = 0.30, 95% CI [-0.21 to 0.80], Standard Error of Mean 0.256
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.5191, Mixed Models Analysis; Mean Difference (Final Values) = 0.16, 95% CI [-0.33 to 0.66], Standard Error of Mean 0.252
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0817, Mixed Models Analysis; Mean Difference (Final Values) = 0.46, 95% CI [-0.06 to 0.97], Standard Error of Mean 0.262
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.1146, Mixed Models Analysis; Mean Difference (Final Values) = 0.40, 95% CI [-0.10 to 0.90], Standard Error of Mean 0.253
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0054, Mixed Models Analysis; Mean Difference (Final Values) = 0.71, 95% CI [0.21 to 1.21], Standard Error of Mean 0.253
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; Week 3: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score is included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.3389, Mixed Models Analysis; Mean Difference (Final Values) = 0.25, 95% CI [-0.26 to 0.76], Standard Error of Mean 0.261
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.5079, Mixed Models Analysis; Mean Difference (Final Values) = 0.17, 95% CI [-0.33 to 0.67], Standard Error of Mean 0.254
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.0453, Mixed Models Analysis; Mean Difference (Final Values) = 0.53, 95% CI [0.01 to 1.05], Standard Error of Mean 0.265
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.1622, Mixed Models Analysis; Mean Difference (Final Values) = 0.36, 95% CI [-0.15 to 0.86], Standard Error of Mean 0.256
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = 0.96, 95% CI [0.45 to 1.48], Standard Error of Mean 0.262
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; Week 4: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score is included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.0383, Mixed Models Analysis; Mean Difference (Final Values) = 0.54, 95% CI [0.03 to 1.05], Standard Error of Mean 0.260
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.4495, Mixed Models Analysis; Mean Difference (Final Values) = 0.19, 95% CI [-0.31 to 0.69], Standard Error of Mean 0.253
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0135, Mixed Models Analysis; Mean Difference (Final Values) = 0.65, 95% CI [0.14 to 1.17], Standard Error of Mean 0.263
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.1423, Mixed Models Analysis; Mean Difference (Final Values) = 0.37, 95% CI [-0.13 to 0.87], Standard Error of Mean 0.254
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0035, Mixed Models Analysis; Mean Difference (Final Values) = 0.76, 95% CI [0.25 to 1.27], Standard Error of Mean 0.259
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 50 mg; Week 5: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score is included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.0125, Mixed Models Analysis; Mean Difference (Final Values) = 0.66, 95% CI [0.14 to 1.17], Standard Error of Mean 0.261
Statistical Analysis 22: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.8021, Mixed Models Analysis; Mean Difference (Final Values) = 0.06, 95% CI [-0.44 to 0.56], Standard Error of Mean 0.254
Statistical Analysis 23: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.0249, Mixed Models Analysis; Mean Difference (Final Values) = 0.60, 95% CI [0.08 to 1.13], Standard Error of Mean 0.267
Statistical Analysis 24: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.3383, Mixed Models Analysis; Mean Difference (Final Values) = 0.25, 95% CI [-0.26 to 0.75], Standard Error of Mean 0.256
Statistical Analysis 25: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.06, 95% CI [0.55 to 1.57], Standard Error of Mean 0.260
Statistical Analysis 26: Comparison: Placebo vs Pregabalin 50 mg; Week 6: Contrast of treatment vs. placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score is included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.0133, Mixed Models Analysis; Mean Difference (Final Values) = 0.65, 95% CI [0.14 to 1.17], Standard Error of Mean 0.261
Statistical Analysis 27: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.3820, Mixed Models Analysis; Mean Difference (Final Values) = 0.22, 95% CI [-0.28 to 0.73], Standard Error of Mean 0.256
Statistical Analysis 28: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0053, Mixed Models Analysis; Mean Difference (Final Values) = 0.75, 95% CI [0.23 to 1.28], Standard Error of Mean 0.269
Statistical Analysis 29: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.3258, Mixed Models Analysis; Mean Difference (Final Values) = 0.25, 95% CI [-0.25 to 0.76], Standard Error of Mean 0.256
Statistical Analysis 30: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Mean Difference (Final Values) = 0.92, 95% CI [0.41 to 1.43], Standard Error of Mean 0.260

6. Secondary Outcome: Subjective Sleep Questionnaire: Number of Awakenings Subscale; Observed Change From Baseline
Description: Subjective Sleep Questionnaire (SSQ): subject-rated instrument used to assess sleep behavior; measures sleep quantity and quality. Comprised of 5 items yielding 5 subscale scores: latency, hours of sleep, number of awakenings, total wake time after sleep onset, and quality of sleep. Number of awakenings subscale: numerical rating completed by the subject 30 minutes after waking; recall period is the night before. Fewer awakenings reflect better quality of sleep. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
Population: ITT; baseline statistics were calculated only for subjects who had a non-missing change from baseline in at least one post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: awakenings
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
awakenings
  Week 1 | -0.5 (0.21) | -0.9 (0.21) | -1.0 (0.21) | -1.2 (0.21) | -0.7 (0.21) | -0.8 (0.21)
  Week 2 | -0.7 (0.21) | -1.0 (0.22) | -1.3 (0.21) | -1.3 (0.23) | -1.3 (0.21) | -1.1 (0.21)
  Week 3 | -0.7 (0.21) | -1.0 (0.22) | -1.0 (0.21) | -1.3 (0.23) | -1.2 (0.21) | -1.4 (0.22)
  Week 4 | -0.9 (0.21) | -1.1 (0.22) | -1.2 (0.21) | -1.5 (0.23) | -1.1 (0.21) | -1.2 (0.22)
  Week 5 | -0.8 (0.21) | -1.3 (0.22) | -1.0 (0.21) | -1.6 (0.23) | -1.2 (0.21) | -1.5 (0.22)
  Week 6 | -1.0 (0.21) | -1.0 (0.22) | -1.1 (0.21) | -1.5 (0.23) | -1.0 (0.21) | -1.2 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1429, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI [-1.0 to 0.1], Standard Error of Mean 0.30
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0547, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI [-1.2 to 0.0], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0095, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI [-1.4 to -0.2], Standard Error of Mean 0.30
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.3676, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI [-0.9 to 0.3], Standard Error of Mean 0.30
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.2959, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI [-0.9 to 0.3], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.3435, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI [-0.9 to 0.3], Standard Error of Mean 0.30
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0895, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI [-1.1 to 0.1], Standard Error of Mean 0.30
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0844, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI [-1.1 to 0.1], Standard Error of Mean 0.31
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0675, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI [-1.1 to 0.0], Standard Error of Mean 0.30
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.2250, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI [-1.0 to 0.2], Standard Error of Mean 0.30
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.3728, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI [-0.9 to 0.3], Standard Error of Mean 0.31
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.2686, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI [-0.9 to 0.3], Standard Error of Mean 0.30
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.0753, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI [-1.2 to 0.1], Standard Error of Mean 0.31
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.1335, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI [-1.0 to 0.1], Standard Error of Mean 0.30
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.0220, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI [-1.3 to -0.1], Standard Error of Mean 0.31
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.5754, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI [-0.8 to 0.4], Standard Error of Mean 0.31
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.3480, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI [-0.9 to 0.3], Standard Error of Mean 0.30
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0554, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI [-1.2 to 0.0], Standard Error of Mean 0.31
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.4362, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI [-0.8 to 0.4], Standard Error of Mean 0.30
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.3631, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI [-0.9 to 0.3], Standard Error of Mean 0.30
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.1152, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI [-1.1 to 0.1], Standard Error of Mean 0.31
Statistical Analysis 22: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.4741, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI [-0.8 to 0.4], Standard Error of Mean 0.30
Statistical Analysis 23: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.0091, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI [-1.4 to -0.2], Standard Error of Mean 0.31
Statistical Analysis 24: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.1721, Mixed Models Analysis; Mean Difference (Final Values) = -0.4, 95% CI [-1.0 to 0.2], Standard Error of Mean 0.30
Statistical Analysis 25: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.0262, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, 95% CI [-1.3 to -0.1], Standard Error of Mean 0.31
Statistical Analysis 26: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.9505, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI [-0.6 to 0.6], Standard Error of Mean 0.31
Statistical Analysis 27: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.6877, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI [-0.7 to 0.5], Standard Error of Mean 0.30
Statistical Analysis 28: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.1271, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI [-1.1 to 0.1], Standard Error of Mean 0.31
Statistical Analysis 29: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.9136, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI [-0.6 to 0.6], Standard Error of Mean 0.30
Statistical Analysis 30: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.4072, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI [-0.9 to 0.3], Standard Error of Mean 0.31

7. Secondary Outcome: Subjective Sleep Questionnaire: Total Wake Time After Sleep Onset Subscale; Observed Change From Baseline
Description: Subjective Sleep Questionnaire (SSQ): subject-rated instrument used to assess sleep behavior; measures sleep quantity and quality. Comprised of 5 items yielding 5 subscale scores: latency, hours of sleep, number of awakenings, total wake time after sleep onset, and quality of sleep. Total wake time after sleep onset subscale (in minutes): numerical rating completed by the subject 30 minutes after waking; recall period is the night before. Reduction = improvement. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | Pregabalin 50 mg/Day | Pregabalin 100 mg/Day | Pregabalin 150 mg/Day | Pregabalin 300 mg/Day | Pregablin 450 mg/Day
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
minutes
  Week 1 | -23.8 (7.44) | -37.9 (7.66) | -28.5 (7.47) | -29.0 (7.81) | -32.2 (7.58) | -32.6 (7.46)
  Week 2 | -29.5 (7.44) | -47.0 (7.79) | -36.5 (7.55) | -41.9 (8.23) | -39.8 (7.68) | -46.3 (7.57)
  Week 3 | -34.3 (7.62) | -51.4 (8.01) | -32.0 (7.47) | -45.9 (8.23) | -42.3 (7.59) | -42.9 (7.89)
  Week 4 | -30.4 (7.53) | -50.7 (8.01) | -36.5 (7.47) | -46.0 (8.23) | -43.6 (7.68) | -46.8 (7.79)
  Week 5 | -28.7 (7.62) | -55.4 (8.01) | -30.7 (7.47) | -59.6 (8.36) | -42.5 (7.59) | -55.1 (7.79)
  Week 6 | -34.2 (7.62) | -57.0 (7.90) | -34.2 (7.55) | -54.0 (8.49) | -41.1 (7.68) | -55.5 (7.89)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg/Day; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1860, Mixed Models Analysis; Mean Difference (Final Values) = -14.2, 95% CI [-35.2 to 6.9], Standard Error of Mean 10.68
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg/Day; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.6530, Mixed Models Analysis; Mean Difference (Final Values) = -4.7, 95% CI [-25.5 to 16.0], Standard Error of Mean 10.54
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg/Day; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.6263, Mixed Models Analysis; Mean Difference (Final Values) = -5.3, 95% CI [-26.5 to 16.0], Standard Error of Mean 10.79
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg/Day; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.4266, Mixed Models Analysis; Mean Difference (Final Values) = -8.5, 95% CI [-29.4 to 12.5], Standard Error of Mean 10.63
Statistical Analysis 5: Comparison: Placebo vs Pregablin 450 mg/Day; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.4023, Mixed Models Analysis; Mean Difference (Final Values) = -8.8, 95% CI [-29.6 to 11.9], Standard Error of Mean 10.54
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg/Day; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.1041, Mixed Models Analysis; Mean Difference (Final Values) = -17.6, 95% CI [-38.8 to 3.6], Standard Error of Mean 10.77
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg/Day; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.5084, Mixed Models Analysis; Mean Difference (Final Values) = -7.0, 95% CI [-27.9 to 13.8], Standard Error of Mean 10.60
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg/Day; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.2620, Mixed Models Analysis; Mean Difference (Final Values) = -12.5, 95% CI [-34.3 to 9.4], Standard Error of Mean 11.10
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg/Day; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.3347, Mixed Models Analysis; Mean Difference (Final Values) = -10.3, 95% CI [-31.4 to 10.7], Standard Error of Mean 10.70
Statistical Analysis 10: Comparison: Placebo vs Pregablin 450 mg/Day; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.1142, Mixed Models Analysis; Mean Difference (Final Values) = -16.8, 95% CI [-37.7 to 4.1], Standard Error of Mean 10.61
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg/Day; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.1237, Mixed Models Analysis; Mean Difference (Final Values) = -17.1, 95% CI [-38.8 to 4.7], Standard Error of Mean 11.06
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg/Day; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.8302, Mixed Models Analysis; Mean Difference (Final Values) = 2.3, 95% CI [-18.7 to 23.3], Standard Error of Mean 10.67
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg/Day; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.3039, Mixed Models Analysis; Mean Difference (Final Values) = -11.6, 95% CI [-33.6 to 10.5], Standard Error of Mean 11.22
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg/Day; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.4595, Mixed Models Analysis; Mean Difference (Final Values) = -8.0, 95% CI [-29.2 to 13.2], Standard Error of Mean 10.77
Statistical Analysis 15: Comparison: Placebo vs Pregablin 450 mg/Day; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.4338, Mixed Models Analysis; Mean Difference (Final Values) = -8.6, 95% CI [-30.2 to 13.0], Standard Error of Mean 10.97
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg/Day; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0647, Mixed Models Analysis; Mean Difference (Final Values) = -20.4, 95% CI [-42.0 to 1.2], Standard Error of Mean 10.99
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg/Day; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.5651, Mixed Models Analysis; Mean Difference (Final Values) = -6.1, 95% CI [-27.0 to 14.8], Standard Error of Mean 10.61
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg/Day; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.1634, Mixed Models Analysis; Mean Difference (Final Values) = -15.6, 95% CI [-37.6 to 6.4], Standard Error of Mean 11.16
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg/Day; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.2209, Mixed Models Analysis; Mean Difference (Final Values) = -13.2, 95% CI [-34.4 to 8.0], Standard Error of Mean 10.77
Statistical Analysis 20: Comparison: Placebo vs Pregablin 450 mg/Day; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.1293, Mixed Models Analysis; Mean Difference (Final Values) = -16.5, 95% CI [-37.8 to 4.8], Standard Error of Mean 10.84
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 50 mg/Day; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.0161, Mixed Models Analysis; Mean Difference (Final Values) = -26.8, 95% CI [-48.5 to -5.0], Standard Error of Mean 11.06
Statistical Analysis 22: Comparison: Placebo vs Pregabalin 100 mg/Day; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.8506, Mixed Models Analysis; Mean Difference (Final Values) = -2.0, 95% CI [-23.0 to 19.0], Standard Error of Mean 10.67
Statistical Analysis 23: Comparison: Placebo vs Pregabalin 150 mg/Day; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.0067, Mixed Models Analysis; Mean Difference (Final Values) = -30.9, 95% CI [-53.2 to -8.6], Standard Error of Mean 11.31
Statistical Analysis 24: Comparison: Placebo vs Pregabalin 300 mg/Day; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.1997, Mixed Models Analysis; Mean Difference (Final Values) = -13.8, 95% CI [-35.0 to 7.4], Standard Error of Mean 10.76
Statistical Analysis 25: Comparison: Placebo vs Pregablin 450 mg/Day; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.0159, Mixed Models Analysis; Mean Difference (Final Values) = -26.4, 95% CI [-47.9 to -5.0], Standard Error of Mean 10.90
Statistical Analysis 26: Comparison: Placebo vs Pregabalin 50 mg/Day; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0388, Mixed Models Analysis; Mean Difference (Final Values) = -22.8, 95% CI [-44.4 to -1.2], Standard Error of Mean 10.98
Statistical Analysis 27: Comparison: Placebo vs Pregabalin 100 mg/Day; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.9962, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI [-21.2 to 21.1], Standard Error of Mean 10.73
Statistical Analysis 28: Comparison: Placebo vs Pregabalin 150 mg/Day; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0839, Mixed Models Analysis; Mean Difference (Final Values) = -19.8, 95% CI [-42.3 to 2.7], Standard Error of Mean 11.41
Statistical Analysis 29: Comparison: Placebo vs Pregabalin 300 mg/Day; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.5216, Mixed Models Analysis; Mean Difference (Final Values) = -6.9, 95% CI [-28.3 to 14.4], Standard Error of Mean 10.83
Statistical Analysis 30: Comparison: Placebo vs Pregablin 450 mg/Day; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0534, Mixed Models Analysis; Mean Difference (Final Values) = -21.3, 95% CI [-42.9 to 0.3], Standard Error of Mean 10.98

8. Secondary Outcome: Subjective Sleep Questionnaire: Quality of Sleep Subscale; Observed Change From Baseline
Description: Subjective Sleep Questionnaire (SSQ): subject-rated instrument used to assess sleep behavior; measures sleep quantity and quality. Comprised of 5 items yielding 5 subscale scores: latency, hours of sleep, number of awakenings, total wake time after sleep onset, and quality of sleep. Quality of sleep subscale: visual analog scale ranging from 1 (very poor) to 100 (excellent) completed by the subject 30 minutes after waking; recall period is the night before. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
scores on scale
  Week 1 | 5.0 (4.10) | 18.8 (4.21) | 15.2 (4.10) | 15.9 (4.23) | 11.5 (4.16) | 17.2 (4.11)
  Week 2 | 11.3 (4.10) | 23.3 (4.27) | 18.7 (4.13) | 24.2 (4.40) | 23.4 (4.20) | 24.0 (4.16)
  Week 3 | 13.8 (4.17) | 23.0 (4.31) | 18.6 (4.10) | 26.8 (4.40) | 23.6 (4.20) | 25.4 (4.29)
  Week 4 | 13.2 (4.14) | 23.8 (4.31) | 22.0 (4.10) | 28.2 (4.40) | 24.2 (4.20) | 23.8 (4.25)
  Week 5 | 14.7 (4.17) | 28.7 (4.31) | 19.9 (4.10) | 30.9 (4.45) | 26.0 (4.20) | 31.1 (4.25)
  Week 6 | 13.9 (4.17) | 27.6 (4.31) | 23.5 (4.14) | 30.5 (4.50) | 23.1 (4.20) | 28.8 (4.25)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0199, Mixed Models Analysis; Mean Difference (Final Values) = 13.8, 95% CI [2.2 to 25.4], Standard Error of Mean 5.89
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0768, Mixed Models Analysis; Mean Difference (Final Values) = 10.3, 95% CI [-1.1 to 21.7], Standard Error of Mean 5.78
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0642, Mixed Models Analysis; Mean Difference (Final Values) = 11.0, 95% CI [-0.7 to 22.6], Standard Error of Mean 5.91
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.2643, Mixed Models Analysis; Median Difference (Final Values) = 6.6, 95% CI [-5.0 to 18.2], Standard Error of Mean 5.88
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0358, Mixed Models Analysis; Mean Difference (Final Values) = 12.2, 95% CI [0.8 to 23.7], Standard Error of Mean 5.80
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0428, Mixed Models Analysis; Mean Difference (Final Values) = 12.1, 95% CI [0.4 to 23.8], Standard Error of Mean 5.93
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.1993, Mixed Models Analysis; Mean Difference (Final Values) = 7.5, 95% CI [-4.0 to 18.9], Standard Error of Mean 5.81
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0331, Mixed Models Analysis; Mean Difference (Final Values) = 12.9, 95% CI [1.1 to 24.8], Standard Error of Mean 6.04
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0415, Mixed Models Analysis; Mean Difference (Final Values) = 12.1, 95% CI [0.5 to 23.8], Standard Error of Mean 5.91
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0295, Mixed Models Analysis; Mean Difference (Final Values) = 12.8, 95% CI [1.3 to 24.3], Standard Error of Mean 5.83
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.1267, Mixed Models Analysis; Mean Difference (Final Values) = 9.2, 95% CI [-2.6 to 21.1], Standard Error of Mean 6.01
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.4175, Mixed Models Analysis; Mean Difference (Final Values) = 4.7, 95% CI [-6.8 to 16.2], Standard Error of Mean 5.84
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.0342, Mixed Models Analysis; Mean Difference (Final Values) = 13.0, 95% CI [1.0 to 25.0], Standard Error of Mean 6.09
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.1038, Mixed Models Analysis; Mean Difference (Final Values) = 9.7, 95% CI [-2.0 to 21.5], Standard Error of Mean 5.96
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; p = 0.0537, Mixed Models Analysis; Mean Difference (Final Values) = 11.6, 95% CI [-0.2 to 23.4], Standard Error of Mean 5.98
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0772, Mixed Models Analysis; Mean Difference (Final Values) = 10.6, 95% CI [-1.2 to 22.4], Standard Error of Mean 5.99
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.1296, Mixed Models Analysis; Mean Difference (Final Values) = 8.8, 95% CI [-2.6 to 20.3], Standard Error of Mean 5.81
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0140, Mixed Models Analysis; Mean Difference (Final Values) = 15.0, 95% CI [3.1 to 27.0], Standard Error of Mean 6.06
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0642, Mixed Models Analysis; Mean Difference (Final Values) = 11.0, 95% CI [-0.7 to 22.7], Standard Error of Mean 5.93
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0730, Mixed Models Analysis; Mean Difference (Final Values) = 10.7, 95% CI [-1.0 to 22.3], Standard Error of Mean 5.92
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.0215, Mixed Models Analysis; Mean Difference (Final Values) = 13.9, 95% CI [2.1 to 25.8], Standard Error of Mean 6.01
Statistical Analysis 22: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.3785, Mixed Models Analysis; Mean Difference (Final Values) = 5.2, 95% CI [-6.4 to 16.7], Standard Error of Mean 5.84
Statistical Analysis 23: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.0089, Mixed Models Analysis; Mean Difference (Final Values) = 16.1, 95% CI [4.1 to 28.2], Standard Error of Mean 6.12
Statistical Analysis 24: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.0609, Mixed Models Analysis; Mean Difference (Final Values) = 11.2, 95% CI [-0.5 to 23.0], Standard Error of Mean 5.96
Statistical Analysis 25: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.0064, Mixed Models Analysis; Mean Difference (Final Values) = 16.4, 95% CI [4.7 to 28.1], Standard Error of Mean 5.95
Statistical Analysis 26: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0241, Mixed Models Analysis; Mean Difference (Final Values) = 13.7, 95% CI [1.8 to 25.5], Standard Error of Mean 6.01
Statistical Analysis 27: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.1032, Mixed Models Analysis; Mean Difference (Final Values) = 9.6, 95% CI [-2.0 to 21.1], Standard Error of Mean 5.86
Statistical Analysis 28: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0076, Mixed Models Analysis; Mean Difference (Final Values) = 16.6, 95% CI [4.4 to 28.7], Standard Error of Mean 6.16
Statistical Analysis 29: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.1257, Mixed Models Analysis; Mean Difference (Final Values) = 9.2, 95% CI [-2.6 to 20.9], Standard Error of Mean 5.96
Statistical Analysis 30: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0131, Mixed Models Analysis; Mean Difference (Final Values) = 14.9, 95% CI [3.2 to 26.6], Standard Error of Mean 5.95

9. Secondary Outcome: Medical Outcomes Study - Sleep Scale (MOSS-SS): Sleep Disturbance Subscale; Observed Change From Baseline
Description: MOS-SS: subject-rated instrument used to assess the key constructs of sleep quantity and quality over the past week; comprised of 12 items yielding 7 subscale scores and 2 composite index scores. Sleep Disturbance Subscale score (4 items): range 0-100; lower score indicates less disturbance. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6
Population: ITT, Baseline statistics were calculated only for subjects who had non-missing change from baseline at at least one post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
scores on scale
  Week 1 | -9.0 (4.76) | -18.2 (5.05) | -21.1 (4.87) | -23.0 (5.26) | -17.7 (4.93) | -26.3 (4.89)
  Week 2 | -15.7 (4.76) | -25.1 (5.14) | -23.0 (4.81) | -26.1 (5.30) | -35.3 (4.95) | -32.1 (5.02)
  Week 4 | -22.0 (4.81) | -18.5 (5.07) | -28.3 (4.76) | -32.4 (5.30) | -34.2 (4.95) | -37.4 (5.02)
  Week 6 | -19.3 (4.87) | -29.2 (5.14) | -25.3 (4.81) | -33.4 (5.38) | -31.4 (4.95) | -40.2 (5.02)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1824, Mixed Models Analysis; Mean Difference (Final Values) = -9.3, 95% CI [-23.0 to 4.4], Standard Error of Mean 6.94
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0767, Mixed Models Analysis; Mean Difference (Final Values) = -12.1, 95% CI [-25.5 to 1.3], Standard Error of Mean 6.80
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0492, Mixed Models Analysis; Mean Difference (Final Values) = -14.1, 95% CI [-28.1 to -0.1], Standard Error of Mean 7.11
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.2023, Mixed Models Analysis; Mean Difference (Final Values) = -8.7, 95% CI [-22.2 to 4.7], Standard Error of Mean 6.84
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0116, Mixed Models Analysis; Mean Difference (Final Values) = -17.4, 95% CI [-30.9 to -3.9], Standard Error of Mean 6.83
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.1819, Mixed Models Analysis; Mean Difference (Final Values) = -9.4, 95% CI [-23.2 to 4.4], Standard Error of Mean 7.01
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.2806, Mixed Models Analysis; Mean Difference (Final Values) = -7.3, 95% CI [-20.6 to 6.0], Standard Error of Mean 6.76
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.1465, Mixed Models Analysis; Mean Difference (Final Values) = -10.4, 95% CI [-24.4 to 3.7], Standard Error of Mean 7.13
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0046, Mixed Models Analysis; Mean Difference (Final Values) = -19.6, 95% CI [-33.1 to -6.1], Standard Error of Mean 6.85
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0187, Mixed Models Analysis; Mean Difference (Final Values) = -16.4, 95% CI [-30.0 to -2.8], Standard Error of Mean 6.92
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.6128, Mixed Models Analysis; Mean Difference (Final Values) = 3.5, 95% CI [-10.2 to 17.3], Standard Error of Mean 7.00
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.3488, Mixed Models Analysis; Mean Difference (Final Values) = -6.4, 95% CI [-19.7 to 7.0], Standard Error of Mean 6.76
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.1472, Mixed Models Analysis; Mean Difference (Final Values) = -10.4, 95% CI [-24.5 to 3.7], Standard Error of Mean 7.17
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0791, Mixed Models Analysis; Mean Difference (Final Values) = -12.2, 95% CI [-25.7 to 1.4], Standard Error of Mean 6.89
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0282, Mixed Models Analysis; Mean Difference (Final Values) = -15.4, 95% CI [-29.1 to -1.7], Standard Error of Mean 6.97
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.1623, Mixed Models Analysis; Mean Difference (Final Values) = -9.9, 95% CI [-23.9 to 4.0], Standard Error of Mean 7.08
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.3739, Mixed Models Analysis; Mean Difference (Final Values) = -6.1, 95% CI [-19.6 to 7.4], Standard Error of Mean 6.84
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0517, Mixed Models Analysis; Mean Difference (Final Values) = -14.2, 95% CI [-28.5 to 0.1], Standard Error of Mean 7.26
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0815, Mixed Models Analysis; Mean Difference (Final Values) = -12.1, 95% CI [-25.8 to 1.5], Standard Error of Mean 6.92
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0031, Mixed Models Analysis; Mean Difference (Final Values) = -20.9, 95% CI [-34.7 to -7.1], Standard Error of Mean 7.00

10. Secondary Outcome: Medical Outcomes Study - Sleep Scale (MOSS-SS): Snoring Subscale; Observed Change From Baseline
Description: MOS-SS: subject-rated instrument used to assess the key constructs of sleep; assesses sleep quantity and quality over the past week. Comprised of 12 items yielding 7 subscale scores and 2 composite index scores. Snoring Subscale score (1 item): range 0-100, lower score indicates less snoring. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
scores on scale
  Week 1 | -2.4 (5.39) | 5.2 (5.72) | -8.6 (5.53) | 0.7 (6.04) | -2.9 (5.46) | -9.2 (5.54)
  Week 2 | -1.5 (5.39) | -0.8 (5.81) | -11.4 (5.47) | -8.7 (6.16) | -3.3 (5.48) | -12.2 (5.66)
  Week 4 | -3.2 (5.44) | 4.4 (5.75) | -4.0 (5.42) | -7.5 (6.16) | 2.8 (5.48) | -3.5 (5.67)
  Week 6 | -2.1 (5.50) | 2.5 (5.81) | -6.6 (5.47) | -2.0 (6.24) | 1.0 (5.48) | -7.5 (5.67)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.3368, Mixed Models Analysis; Mean Difference (Final Values) = 7.6, 95% CI [-8.0 to 23.1], Standard Error of Mean 7.88
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.4232, Mixed Models Analysis; Mean Difference (Final Values) = -6.2, 95% CI [-21.5 to 9.1], Standard Error of Mean 7.75
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.7082, Mixed Models Analysis; Mean Difference (Final Values) = 3.0, 95% CI [-12.9 to 19.0], Standard Error of Mean 8.09
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.9466, Mixed Models Analysis; Mean Difference (Final Values) = -0.5, 95% CI [-15.7 to 14.7], Standard Error of Mean 7.70
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.3746, Mixed Models Analysis; Mean Difference (Final Values) = -6.9, 95% CI [-22.1 to 8.4], Standard Error of Mean 7.72
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.9336, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI [-15.0 to 16.3], Standard Error of Mean 7.95
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.2029, Mixed Models Analysis; Mean Difference (Final Values) = -9.8, 95% CI [-25.0 to 5.4], Standard Error of Mean 7.71
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.3833, Mixed Models Analysis; Mean Difference (Final Values) = -7.1, 95% CI [-23.3 to 9.0], Standard Error of Mean 8.18
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.8152, Mixed Models Analysis; Mean Difference (Final Values) = -1.8, 95% CI [-17.0 to 13.4], Standard Error of Mean 7.72
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.1739, Mixed Models Analysis; Mean Difference (Final Values) = -10.7, 95% CI [-26.1 to 4.7], Standard Error of Mean 7.81
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.3392, Mixed Models Analysis; Mean Difference (Final Values) = 7.6, 95% CI [-8.0 to 23.3], Standard Error of Mean 7.94
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.9130, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI [-16.0 to 14.4], Standard Error of Mean 7.71
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.6000, Mixed Models Analysis; Mean Difference (Final Values) = -4.3, 95% CI [-20.5 to 11.9], Standard Error of Mean 8.22
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.4445, Mixed Models Analysis; Mean Difference (Final Values) = 5.9, 95% CI [-9.3 to 21.2], Standard Error of Mean 7.75
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.9656, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI [-15.8 to 15.1], Standard Error of Mean 7.85
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.5679, Mixed Models Analysis; Mean Difference (Final Values) = 4.6, 95% CI [-11.2 to 20.4], Standard Error of Mean 8.02
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.5619, Mixed Models Analysis; Mean Difference (Final Values) = -4.5, 95% CI [-19.9 to 10.8], Standard Error of Mean 7.79
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.9930, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI [-16.3 to 16.4], Standard Error of Mean 8.31
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.6892, Mixed Models Analysis; Mean Difference (Final Values) = 3.1, 95% CI [-12.2 to 18.5], Standard Error of Mean 7.79
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.4928, Mixed Models Analysis; Mean Difference (Final Values) = -5.4, 95% CI [-21.0 to 10.1], Standard Error of Mean 7.89

11. Secondary Outcome: Medical Outcomes Study - Sleep Scale (MOSS-SS): Awaken Short of Breath or With Headache Subscale; Observed Change From Baseline
Description: MOS-SS: subject-rated instrument used to assess the key constructs of sleep over the past week ; comprised of 12 items yielding 7 subscale scores and 2 composite index scores. Awaken Short of Breath or with Headache subscale score range: 0-100; lower score indicates less difficulty. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
scores on scale
  Week 1 | -7.3 (3.49) | -1.7 (3.72) | -5.3 (3.62) | -9.2 (3.92) | -8.6 (3.51) | 1.4 (3.58)
  Week 2 | -9.1 (3.49) | -4.3 (3.81) | -8.8 (3.54) | -12.1 (3.93) | -8.2 (3.53) | -1.1 (3.72)
  Week 4 | -9.9 (3.56) | -2.5 (3.73) | -8.9 (3.47) | -9.9 (3.93) | -9.1 (3.53) | -9.2 (3.73)
  Week 6 | -7.4 (3.63) | -0.9 (3.81) | -4.9 (3.54) | -11.5 (4.03) | -3.0 (3.53) | -8.2 (3.73)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; Week 1: Contrast of treatment vs placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score is included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.2719, Mixed Models Analysis; Mean Difference (Final Values) = 5.6, 95% CI [-4.4 to 15.6], Standard Error of Mean 5.10
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.6930, Mixed Models Analysis; Mean Difference (Final Values) = 2.0, 95% CI [-7.9 to 11.8], Standard Error of Mean 5.02
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.7178, Mixed Models Analysis; Mean Difference (Final Values) = -1.9, 95% CI [-12.2 to 8.4], Standard Error of Mean 5.24
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.8037, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI [-11.0 to 8.5], Standard Error of Mean 4.96
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.0832, Mixed Models Analysis; Mean Difference (Final Values) = 8.7, 95% CI [-1.2 to 18.6], Standard Error of Mean 5.02
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; Week 2: Contrast of treatment vs placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score is included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.3554, Mixed Models Analysis; Mean Difference (Final Values) = 4.8, 95% CI [-5.4 to 14.9], Standard Error of Mean 5.17
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.9538, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI [-9.5 to 10.0], Standard Error of Mean 4.96
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.5593, Mixed Models Analysis; Mean Difference (Final Values) = -3.1, 95% CI [-13.4 to 7.3], Standard Error of Mean 5.26
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.8663, Mixed Models Analysis; Mean Difference (Final Values) = 0.8, 95% CI [-8.9 to 10.6], Standard Error of Mean 4.97
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.1190, Mixed Models Analysis; Mean Difference (Final Values) = 8.0, 95% CI [-2.1 to 18.1], Standard Error of Mean 5.12
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; Week 4: Contrast of treatment vs placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score is included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.1544, Mixed Models Analysis; Mean Difference (Final Values) = 7.4, 95% CI [-2.8 to 17.5], Standard Error of Mean 5.15
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.8439, Mixed Models Analysis; Mean Difference (Final Values) = 1.0, 95% CI [-8.8 to 10.7], Standard Error of Mean 4.97
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.9925, Mixed Models Analysis; Mean Difference (Final Values) = -0.0, 95% CI [-10.5 to 10.4], Standard Error of Mean 5.30
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.8784, Mixed Models Analysis; Mean Difference (Final Values) = 0.8, 95% CI [-9.1 to 10.6], Standard Error of Mean 5.02
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.8948, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI [-9.5 to 10.8], Standard Error of Mean 5.17
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; Week 6: Contrast of treatment vs placebo. Repeated measures model used fixed effects of treatment, geographic region, week and treatment by week interaction. Baseline score is included as a covariate. Additionally, the model includes subject as a repeated measurement block within which the covariance structure is assumed to be compound symmetric (CS); Test type: Superiority or Other; p = 0.2197, Mixed Models Analysis; Mean Difference (Final Values) = 6.5, 95% CI [-3.9 to 16.8], Standard Error of Mean 5.26
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.6183, Mixed Models Analysis; Mean Difference (Final Values) = 2.5, 95% CI [-7.4 to 12.5], Standard Error of Mean 5.07
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.4484, Mixed Models Analysis; Mean Difference (Final Values) = -4.1, 95% CI [-14.8 to 6.5], Standard Error of Mean 5.42
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.3857, Mixed Models Analysis; Mean Difference (Final Values) = 4.4, 95% CI [-5.6 to 14.4], Standard Error of Mean 5.07
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.8824, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI [-11.0 to 9.5], Standard Error of Mean 5.22

12. Secondary Outcome: Medical Outcomes Study - Sleep Scale (MOSS-SS): Sleep Adequacy Subscale; Observed Change From Baseline
Description: MOS-SS: subject-rated instrument used to assess the key constructs of sleep; assesses sleep quantity and quality and is comprised 12 items yielding 7 subscale scores and 2 composite index scores. Sleep Adequacy Subscale score range: 0-100; higher scores indicates greater sleep adequacy. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
scores on scale
  Week 1 | 5.2 (5.38) | 16.1 (5.76) | 5.3 (5.53) | 13.7 (6.01) | 9.8 (5.50) | 16.1 (5.58)
  Week 2 | 15.6 (5.38) | 31.0 (5.87) | 19.6 (5.45) | 21.9 (6.06) | 14.0 (5.53) | 29.5 (5.76)
  Week 4 | 15.6 (5.45) | 23.9 (5.78) | 20.8 (5.38) | 24.7 (6.06) | 26.6 (5.53) | 34.6 (5.78)
  Week 6 | 16.8 (5.54) | 34.6 (5.87) | 27.0 (5.45) | 26.8 (6.17) | 19.2 (5.53) | 31.1 (5.78)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1673, Mixed Models Analysis; Mean Difference (Final Values) = 10.9, 95% CI [-4.6 to 26.4], Standard Error of Mean 7.87
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.9839, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI [-15.0 to 15.3], Standard Error of Mean 7.71
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.2905, Mixed Models Analysis; Mean Difference (Final Values) = 8.5, 95% CI [-7.3 to 24.4], Standard Error of Mean 8.06
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.5513, Mixed Models Analysis; Mean Difference (Final Values) = 4.6, 95% CI [-10.6 to 19.7], Standard Error of Mean 7.69
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1589, Mixed Models Analysis; Mean Difference (Final Values) = 11.0, 95% CI [-4.3 to 26.3], Standard Error of Mean 7.77
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0541, Mixed Models Analysis; Mean Difference (Final Values) = 15.4, 95% CI [-0.3 to 31.0], Standard Error of Mean 7.95
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.5987, Mixed Models Analysis; Mean Difference (Final Values) = 4.0, 95% CI [-11.0 to 19.1], Standard Error of Mean 7.66
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.4372, Mixed Models Analysis; Mean Difference (Final Values) = 6.3, 95% CI [-9.6 to 22.2], Standard Error of Mean 8.10
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.8336, Mixed Models Analysis; Mean Difference (Final Values) = -1.6, 95% CI [-16.8 to 13.6], Standard Error of Mean 7.71
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0804, Mixed Models Analysis; Mean Difference (Final Values) = 13.9, 95% CI [-1.7 to 29.4], Standard Error of Mean 7.90
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.2985, Mixed Models Analysis; Mean Difference (Final Values) = 8.3, 95% CI [-7.4 to 23.9], Standard Error of Mean 7.94
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.4991, Mixed Models Analysis; Mean Difference (Final Values) = 5.2, 95% CI [-9.9 to 20.3], Standard Error of Mean 7.66
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.2675, Mixed Models Analysis; Mean Difference (Final Values) = 9.1, 95% CI [-7.0 to 25.1], Standard Error of Mean 8.15
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.1593, Mixed Models Analysis; Mean Difference (Final Values) = 11.0, 95% CI [-4.3 to 26.3], Standard Error of Mean 7.77
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0179, Mixed Models Analysis; Mean Difference (Final Values) = 18.9, 95% CI [3.3 to 34.6], Standard Error of Mean 7.96
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0281, Mixed Models Analysis; Mean Difference (Final Values) = 17.8, 95% CI [1.9 to 33.7], Standard Error of Mean 8.06
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.1883, Mixed Models Analysis; Mean Difference (Final Values) = 10.3, 95% CI [-5.0 to 25.5], Standard Error of Mean 7.77
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.2300, Mixed Models Analysis; Mean Difference (Final Values) = 10.0, 95% CI [-6.3 to 26.3], Standard Error of Mean 8.28
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.7575, Mixed Models Analysis; Mean Difference (Final Values) = 2.4, 95% CI [-13.0 to 17.8], Standard Error of Mean 7.82
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0757, Mixed Models Analysis; Mean Difference (Final Values) = 14.3, 95% CI [-1.5 to 30.1], Standard Error of Mean 8.02

13. Secondary Outcome: Medical Outcomes Study - Sleep Scale (MOSS-SS): Somnolence Subscale; Observed Change From Baseline
Description: MOS-SS: subject-rated instrument used to assess the key constructs of sleep over the past week; assesses sleep quantity and quality and is comprised 12 items yielding 7 subscale scores and 2 composite index scores. Sleep Somnolence Subscale score range: 0-100; higher score indicates less somnolence. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline,, Week 1, Week 2, Week 4, Week 6
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
scores on scale
  Week 1 | -7.4 (4.02) | -13.8 (4.29) | -9.8 (4.12) | -14.3 (4.46) | -11.2 (4.07) | -10.7 (4.14)
  Week 2 | -13.9 (4.02) | -18.2 (4.36) | -11.1 (4.07) | -18.8 (4.49) | -11.3 (4.09) | -12.6 (4.25)
  Week 4 | -14.0 (4.07) | -20.4 (4.30) | -11.8 (4.02) | -16.2 (4.49) | -16.9 (4.09) | -12.6 (4.26)
  Week 6 | -11.7 (4.12) | -26.3 (4.36) | -14.8 (4.07) | -21.7 (4.56) | -13.4 (4.09) | -13.9 (4.26)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.2817, Mixed Models Analysis; Mean Difference (Final Values) = -6.4, 95% CI [-18.0 to 5.2], Standard Error of Mean 5.89
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.6796, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI [-13.7 to 9.0], Standard Error of Mean 5.76
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.2505, Mixed Models Analysis; Mean Difference (Final Values) = -6.9, 95% CI [-18.8 to 4.9], Standard Error of Mean 6.01
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.5102, Mixed Models Analysis; Mean Difference (Final Values) = -3.8, 95% CI [-15.1 to 7.5], Standard Error of Mean 5.73
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.5706, Mixed Models Analysis; Mean Difference (Final Values) = -3.3, 95% CI [-14.7 to 8.1], Standard Error of Mean 5.78
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.4708, Mixed Models Analysis; Mean Difference (Final Values) = -4.3, 95% CI [-16.0 to 7.4], Standard Error of Mean 5.95
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.6202, Mixed Models Analysis; Mean Difference (Final Values) = 2.8, 95% CI [-8.4 to 14.1], Standard Error of Mean 5.72
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.4177, Mixed Models Analysis; Mean Difference (Final Values) = -4.9, 95% CI [-16.8 to 7.0], Standard Error of Mean 6.04
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.6509, Mixed Models Analysis; Mean Difference (Final Values) = 2.6, 95% CI [-8.7 to 13.9], Standard Error of Mean 5.75
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.8273, Mixed Models Analysis; Mean Difference (Final Values) = 1.3, 95% CI [-10.3 to 12.8], Standard Error of Mean 5.86
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.2842, Mixed Models Analysis; Mean Difference (Final Values) = -6.4, 95% CI [-18.1 to 5.3], Standard Error of Mean 5.94
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.7041, Mixed Models Analysis; Mean Difference (Final Values) = 2.2, 95% CI [-9.1 to 13.5], Standard Error of Mean 5.72
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.7216, Mixed Models Analysis; Mean Difference (Final Values) = -2.2, 95% CI [-14.1 to 9.8], Standard Error of Mean 6.07
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.6188, Mixed Models Analysis; Mean Difference (Final Values) = -2.9, 95% CI [-14.3 to 8.5], Standard Error of Mean 5.78
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.8096, Mixed Models Analysis; Mean Difference (Final Values) = 1.4, 95% CI [-10.2 to 13.0], Standard Error of Mean 5.90
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.0157, Mixed Models Analysis; Mean Difference (Final Values) = -14.6, 95% CI [-26.5 to -2.8], Standard Error of Mean 6.01
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.6007, Mixed Models Analysis; Mean Difference (Final Values) = -3.0, 95% CI [-14.4 to 8.4], Standard Error of Mean 5.79
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.1057, Mixed Models Analysis; Mean Difference (Final Values) = -10.0, 95% CI [-22.1 to 2.1], Standard Error of Mean 6.15
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.7764, Mixed Models Analysis; Mean Difference (Final Values) = -1.7, 95% CI [-13.1 to 9.8], Standard Error of Mean 5.81
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.7146, Mixed Models Analysis; Mean Difference (Final Values) = -2.2, 95% CI [-13.9 to 9.5], Standard Error of Mean 5.93

14. Secondary Outcome: Medical Outcomes Study - Sleep Scale (MOSS-SS): Sleep Quantity Subscale; Observed Change From Baseline
Description: MOS-SS: subject-rated instrument used to assess the key constructs of sleep over the past week; assesses sleep quantity and quality and is comprised 12 items yielding 7 subscale scores and 2 composite index scores. Sleep Quantity (1 item) subscale score range: 0-24 hours. Change from Baseline in number of hours slept. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline,, Week 1, Week 2, Week 4, Week 6
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
scores on scale
  Week 1 | 0.4 (0.21) | 0.7 (0.22) | 0.5 (0.22) | 0.9 (0.23) | 0.4 (0.21) | 0.7 (0.22)
  Week 2 | 0.5 (0.21) | 0.8 (0.23) | 0.6 (0.21) | 1.2 (0.23) | 0.7 (0.21) | 1.1 (0.22)
  Week 4 | 0.6 (0.21) | 1.0 (0.22) | 0.7 (0.21) | 1.4 (0.23) | 1.1 (0.21) | 1.1 (0.22)
  Week 6 | 0.6 (0.22) | 0.9 (0.23) | 0.7 (0.21) | 1.3 (0.24) | 0.7 (0.21) | 1.2 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.2978, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI [-0.3 to 0.9], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.7242, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI [-0.5 to 0.7], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0773, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI [-0.1 to 1.2], Standard Error of Mean 0.32
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.7831, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI [-0.5 to 0.7], Standard Error of Mean 0.30
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.3291, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI [-0.3 to 0.9], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.3692, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI [-0.3 to 0.9], Standard Error of Mean 0.31
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.7614, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI [-0.5 to 0.7], Standard Error of Mean 0.30
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0355, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI [0.0 to 1.3], Standard Error of Mean 0.32
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.5068, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI [-0.4 to 0.8], Standard Error of Mean 0.30
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0561, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI [-0.0 to 1.2], Standard Error of Mean 0.31
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.2223, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI [-0.2 to 1.0], Standard Error of Mean 0.31
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.6791, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI [-0.5 to 0.7], Standard Error of Mean 0.30
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0188, Mixed Models Analysis; Mean Difference (Final Values) = 0.8, 95% CI [0.1 to 1.4], Standard Error of Mean 0.32
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.1314, Mixed Models Analysis; Mean Difference (Final Values) = 0.5, 95% CI [-0.1 to 1.1], Standard Error of Mean 0.30
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0900, Mixed Models Analysis; Mean Difference (Final Values) = 0.5, 95% CI [-0.1 to 1.1], Standard Error of Mean 0.31
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.4144, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI [-0.4 to 0.9], Standard Error of Mean 0.31
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.7699, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI [-0.5 to 0.7], Standard Error of Mean 0.30
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0406, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI [0.0 to 1.3], Standard Error of Mean 0.32
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.7574, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI [-0.5 to 0.7], Standard Error of Mean 0.30
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0554, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI [-0.0 to 1.2], Standard Error of Mean 0.31

15. Secondary Outcome: Medical Outcomes Study - Sleep Scale (MOSS-SS): 6-Item Sleep Problems Index; Observed Change From Baseline
Description: MOS-SS: subject-rated instrument used to assess the key constructs of sleep over the past week; assesses sleep quantity and quality and is comprised 12 items yielding 7 subscale scores and 2 composite index scores. Sleep Problems Index I (6 items): composite index score range 0-100; lower score indicates fewer sleep problems. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
scores on scale
  Week 1 | -9.2 (3.67) | -12.5 (3.91) | -10.4 (3.75) | -14.9 (4.06) | -13.9 (3.77) | -16.2 (3.77)
  Week 2 | -14.8 (3.67) | -22.0 (3.97) | -15.7 (3.71) | -20.3 (4.09) | -20.1 (3.79) | -24.1 (3.87)
  Week 4 | -17.2 (3.71) | -17.9 (3.92) | -19.6 (3.67) | -23.3 (4.09) | -24.4 (3.79) | -28.9 (3.88)
  Week 6 | -15.5 (3.76) | -25.0 (3.97) | -21.1 (3.71) | -26.1 (4.15) | -18.8 (3.79) | -27.6 (3.88)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.5409, Mixed Models Analysis; Mean Difference (Final Values) = -3.3, 95% CI [-13.8 to 7.3], Standard Error of Mean 5.36
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.8230, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI [-11.5 to 9.2], Standard Error of Mean 5.25
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.2958, Mixed Models Analysis; Mean Difference (Final Values) = -5.7, 95% CI [-16.5 to 5.1], Standard Error of Mean 5.48
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.3708, Mixed Models Analysis; Mean Difference (Final Values) = -4.7, 95% CI [-15.1 to 5.7], Standard Error of Mean 5.27
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1853, Mixed Models Analysis; Mean Difference (Final Values) = -7.0, 95% CI [-17.4 to 3.4], Standard Error of Mean 5.27
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.1834, Mixed Models Analysis; Mean Difference (Final Values) = -7.2, 95% CI [-17.9 to 3.4], Standard Error of Mean 5.41
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.8711, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI [-11.1 to 9.4], Standard Error of Mean 5.22
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.3252, Mixed Models Analysis; Mean Difference (Final Values) = -5.4, 95% CI [-16.3 to 5.4], Standard Error of Mean 5.50
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.3205, Mixed Models Analysis; Mean Difference (Final Values) = -5.3, 95% CI [-15.7 to 5.1], Standard Error of Mean 5.28
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.0837, Mixed Models Analysis; Mean Difference (Final Values) = -9.3, 95% CI [-19.8 to 1.2], Standard Error of Mean 5.34
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.8895, Mixed Models Analysis; Mean Difference (Final Values) = -0.8, 95% CI [-11.4 to 9.9], Standard Error of Mean 5.40
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.6469, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI [-12.7 to 7.9], Standard Error of Mean 5.22
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.2687, Mixed Models Analysis; Mean Difference (Final Values) = -6.1, 95% CI [-17.0 to 4.8], Standard Error of Mean 5.53
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.1757, Mixed Models Analysis; Mean Difference (Final Values) = -7.2, 95% CI [-17.7 to 3.3], Standard Error of Mean 5.31
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 16]; Test type: Superiority or Other; p = 0.0306, Mixed Models Analysis; Mean Difference (Final Values) = -11.7, 95% CI [-22.3 to -1.1], Standard Error of Mean 5.38
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0857, Mixed Models Analysis; Mean Difference (Final Values) = -9.4, 95% CI [-20.2 to 1.3], Standard Error of Mean 5.47
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.2932, Mixed Models Analysis; Mean Difference (Final Values) = -5.6, 95% CI [-16.0 to 4.8], Standard Error of Mean 5.28
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0613, Mixed Models Analysis; Mean Difference (Final Values) = -10.5, 95% CI [-21.6 to 0.5], Standard Error of Mean 5.60
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.5431, Mixed Models Analysis; Mean Difference (Final Values) = -3.3, 95% CI [-13.8 to 7.3], Standard Error of Mean 5.34
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 5, analysis 26]; Test type: Superiority or Other; p = 0.0262, Mixed Models Analysis; Mean Difference (Final Values) = -12.1, 95% CI [-22.7 to -1.4], Standard Error of Mean 5.41

16. Secondary Outcome: Medical Outcomes Study - Sleep Scale (MOSS-SS): 9-Item Sleep Problems Index; Observed Change From Baseline
Description: MOS-SS: subject-rated instrument used to assess the key constructs of sleep over the past week; assesses sleep quantity and quality and is comprised 12 items yielding 7 subscale scores and 2 composite index scores. Composite index scores are sleep problems Index I (6 items) and sleep problems Index II (9 items). 9-Item Sleep Problems Index range: 0-100; lower score indicates fewer sleep problems. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
scores on scale
  Week 1 | -8.1 (3.73) | -15.9 (3.96) | -14.2 (3.81) | -17.8 (4.12) | -14.4 (3.84) | -18.8 (3.83)
  Week 2 | -15.5 (3.73) | -23.5 (4.03) | -19.0 (3.76) | -22.5 (4.15) | -23.3 (3.86) | -24.6 (3.93)
  Week 4 | -18.2 (3.77) | -19.3 (3.98) | -22.0 (3.73) | -25.2 (4.15) | -27.0 (3.86) | -29.1 (3.93)
  Week 6 | -16.8 (3.81) | -27.5 (4.03) | -22.2 (3.76) | -28.3 (4.21) | -22.3 (3.86) | -29.4 (3.93)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.1547, Mixed Models Analysis; Mean Difference (Final Values) = -7.8, 95% CI [-18.5 to 3.0], Standard Error of Mean 5.44
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.2532, Mixed Models Analysis; Mean Difference (Final Values) = -6.1, 95% CI [-16.6 to 4.4], Standard Error of Mean 5.33
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.0848, Mixed Models Analysis; Mean Difference (Final Values) = -9.6, 95% CI [-20.6 to 1.3], Standard Error of Mean 5.56
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.2424, Mixed Models Analysis; Mean Difference (Final Values) = -6.3, 95% CI [-16.8 to 4.3], Standard Error of Mean 5.36
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.0470, Mixed Models Analysis; Mean Difference (Final Values) = -10.7, 95% CI [-21.2 to -0.1], Standard Error of Mean 5.35
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.1494, Mixed Models Analysis; Mean Difference (Final Values) = -7.9, 95% CI [-18.8 to 2.9], Standard Error of Mean 5.49
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.5081, Mixed Models Analysis; Mean Difference (Final Values) = -3.5, 95% CI [-13.9 to 6.9], Standard Error of Mean 5.30
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.2141, Mixed Models Analysis; Mean Difference (Final Values) = -7.0, 95% CI [-17.9 to 4.0], Standard Error of Mean 5.58
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.1484, Mixed Models Analysis; Mean Difference (Final Values) = -7.8, 95% CI [-18.4 to 2.8], Standard Error of Mean 5.37
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.0963, Mixed Models Analysis; Mean Difference (Final Values) = -9.0, 95% CI [-19.7 to 1.6], Standard Error of Mean 5.42
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.8519, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI [-11.8 to 9.8], Standard Error of Mean 5.48
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.4770, Mixed Models Analysis; Mean Difference (Final Values) = -3.8, 95% CI [-14.2 to 6.7], Standard Error of Mean 5.30
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.2166, Mixed Models Analysis; Mean Difference (Final Values) = -6.9, 95% CI [-18.0 to 4.1], Standard Error of Mean 5.61
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.1062, Mixed Models Analysis; Mean Difference (Final Values) = -8.8, 95% CI [-19.4 to 1.9], Standard Error of Mean 5.40
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.0475, Mixed Models Analysis; Mean Difference (Final Values) = -10.9, 95% CI [-21.6 to -0.1], Standard Error of Mean 5.45
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.0537, Mixed Models Analysis; Mean Difference (Final Values) = -10.7, 95% CI [-21.7 to 0.2], Standard Error of Mean 5.54
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.3153, Mixed Models Analysis; Mean Difference (Final Values) = -5.4, 95% CI [-15.9 to 5.2], Standard Error of Mean 5.35
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.0424, Mixed Models Analysis; Mean Difference (Final Values) = -11.6, 95% CI [-22.8 to -0.4], Standard Error of Mean 5.68
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.3077, Mixed Models Analysis; Mean Difference (Final Values) = -5.5, 95% CI [-16.2 to 5.1], Standard Error of Mean 5.42
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 11, analysis 16]; Test type: Superiority or Other; p = 0.0224, Mixed Models Analysis; Mean Difference (Final Values) = -12.6, 95% CI [-23.4 to -1.8], Standard Error of Mean 5.48

17. Secondary Outcome: Medical Outcomes Study - Sleep Scale (MOSS-SS): Optimal Sleep; Observed Cases Summarized by Week
Description: MOS-SS: subject-rated instrument used to assess the key constructs of sleep over the past week; assesses sleep quantity and quality and is comprised 12 items yielding 7 subscale scores and 2 composite index scores. Optimal Sleep subscale is derived from sleep quantity average hours of sleep each night during the past week. Number of subjects with response: YES (Optimal) if sleep quantity was 7 or 8 hours of sleep per night.
Time Frame: Week 1, Week 2, Week 4, Week 6
Population: ITT
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
participants
  Week 1 | 6 | 10 | 7 | 9 | 6 | 11
  Week 2 | 8 | 6 | 11 | 9 | 12 | 12
  Week 4 | 11 | 12 | 11 | 10 | 14 | 11
  Week 6 | 12 | 11 | 11 | 10 | 9 | 13
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; Week 1: Contrast of treatment vs. placebo. Differences in proportions were obtained using LS means. Repeated measures logistic regression model used fixed effects including treatment, geographic region, week, and the treatment by week interaction. The within-subject covariance structure was modeled as compound sysmetric; Test type: Superiority or Other; p = 0.0646, Regression, Logistic; Odds Ratio (OR) = 3.7, 95% CI [0.9 to 15.0], Standard Error of Mean 2.65
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.2947, Regression, Logistic; Odds Ratio (OR) = 2.2, 95% CI [0.5 to 9.1], Standard Error of Mean 1.58
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.0249, Regression, Logistic; Odds Ratio (OR) = 4.6, 95% CI [1.2 to 17.2], Standard Error of Mean 3.10
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.7671, Regression, Logistic; Odds Ratio (OR) = 1.3, 95% CI [0.3 to 5.9], Standard Error of Mean 0.99
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.0169, Regression, Logistic; Odds Ratio (OR) = 4.6, 95% CI [1.3 to 15.9], Standard Error of Mean 2.90
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; Week 2: Contrast of treatment vs. placebo. Differences in proportions were obtained using LS means. Repeated measures logistic regression model used fixed effects including treatment, geographic region, week, and the treatment by week interaction. The within-subject covariance structure was modeled as compound sysmetric; Test type: Superiority or Other; p = 0.9569, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI [0.2 to 4.3], Standard Error of Mean 0.74
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; Week 2: Contrast of treatment vs. placebo. Differences in proportions were obtained using LS means.Repeated measures logistic regression model used fixed effects including treatment, geographic region, week, and the treatment by week interaction. The within-subject covariance structure was modeled as compound sysmetric; Test type: Superiority or Other; p = 0.0711, Regression, Logistic; Odds Ratio (OR) = 3.2, 95% CI [0.9 to 11.4], Standard Error of Mean 2.07
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 17, analysis 6]; Test type: Superiority or Other; p = 0.1073, Regression, Logistic; Odds Ratio (OR) = 2.8, 95% CI [0.8 to 10.2], Standard Error of Mean 1.85
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 17, analysis 6]; Test type: Superiority or Other; p = 0.1583, Regression, Logistic; Odds Ratio (OR) = 2.4, 95% CI [0.7 to 8.1], Standard Error of Mean 1.48
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 17, analysis 6]; Test type: Superiority or Other; p = 0.0385, Regression, Logistic; Odds Ratio (OR) = 4.1, 95% CI [1.1 to 15.6], Standard Error of Mean 2.80
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; Week 4: Contrast of treatment vs. placebo. Differences in proportions were obtained using LS means. Repeated measures logistic regression model used fixed effects including treatment, geographic region, week, and the treatment by week interaction. The within-subject covariance structure was modeled as compound sysmetric; Test type: Superiority or Other; p = 0.4923, Regression, Logistic; Odds Ratio (OR) = 1.6, 95% CI [0.4 to 6.1], Standard Error of Mean 1.09
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 17, analysis 11]; Test type: Superiority or Other; p = 0.7169, Regression, Logistic; Odds Ratio (OR) = 1.3, 95% CI [0.4 to 4.4], Standard Error of Mean 0.80
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 17, analysis 11]; Test type: Superiority or Other; p = 0.4156, Regression, Logistic; Odds Ratio (OR) = 1.7, 95% CI [0.5 to 6.2], Standard Error of Mean 1.12
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 17, analysis 11]; Test type: Superiority or Other; p = 0.4165, Regression, Logistic; Odds Ratio (OR) = 1.7, 95% CI [0.5 to 5.6], Standard Error of Mean 1.04
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 17, analysis 11]; Test type: Superiority or Other; p = 0.4673, Regression, Logistic; Odds Ratio (OR) = 1.6, 95% CI [0.4 to 6.0], Standard Error of Mean 1.08
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; Week 6: Contrast of treatment vs. placebo. Differences in proportions were obtained using LS means. Repeated measures logistic regression model used fixed effects including treatment, geographic region, week, and the treatment by week interaction. The within-subject covariance structure was modeled as compound sysmetric; Test type: Superiority or Other; p = 0.9855, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI [0.2 to 4.1], Standard Error of Mean 0.72
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 17, analysis 16]; Test type: Superiority or Other; p = 0.9566, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI [0.3 to 3.3], Standard Error of Mean 0.61
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 17, analysis 16]; Test type: Superiority or Other; p = 0.4632, Regression, Logistic; Odds Ratio (OR) = 1.7, 95% CI [0.4 to 6.6], Standard Error of Mean 1.17
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 17, analysis 16]; Test type: Superiority or Other; p = 0.2042, Regression, Logistic; Odds Ratio (OR) = 0.4, 95% CI [0.1 to 1.6], Standard Error of Mean 0.29
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 17, analysis 16]; Test type: Superiority or Other; p = 0.3382, Regression, Logistic; Odds Ratio (OR) = 1.9, 95% CI [0.5 to 7.5], Standard Error of Mean 1.34

18. Secondary Outcome: Restless Leg Syndrome - Quality of Life Scale (RLS-QoL): Change From Baseline to Week 6
Description: RLS QoL: subject-rated instrument used to assess the impact of RLS on quality of life and health status function (symptom severity, daily activity, social functioning, sleep, concentrating and decision making, traveling, sexual activity, and work) yielding a summary score ranging from 0-100. Higher scores reflect better quality of life. Recall period is the month prior to the assessment. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 6
Population: ITT; N = Subjects who were randomized and received at least one dose of study drug; baseline n = subjects who were randomized and received at least one dose of study drug, and had baseline and post-baseline values.
Measure: Least Squares Mean (Standard Error); unit: scores on scales
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
scores on scales | 15.0 (3.71) | 19.6 (3.87) | 22.4 (3.55) | 20.8 (3.94) | 15.9 (3.63) | 20.5 (3.74)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; Analysis of covariance of change from baseline; LS Mean, standard error, 95% CI and P-value are from an analysis of covariance (ANCOVA), with treatment and geographic region as main effects and baseline value as covariate in the model; Test type: Superiority or Other; p = 0.3932, ANCOVA; Mean Difference (Final Values) = 4.6, 95% CI [-6.0 to 15.2]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.1585, ANCOVA; Mean Difference (Final Values) = 7.3, 95% CI [-2.9 to 17.5]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.2850, ANCOVA; Mean Difference (Final Values) = 5.8, 95% CI [-4.9 to 16.5]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.8645, ANCOVA; Mean Difference (Final Values) = 0.9, 95% CI [-9.4 to 11.1]
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.3031, ANCOVA; Mean Difference (Final Values) = 5.4, 95% CI [-5.0 to 15.8]

19. Secondary Outcome: Medical Outcomes Study Short Form 36 (SF-36): Change From Baseline to Week 6
Description: Subject-rated measure of health status comprised of 36 items: 8 subscale scores (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health), 2 summary scores (physical component and mental component), and a self-evaluated change in health status. Subscale and summary scores range: 0-100. Higher subscale and summary scores = better health status. Recall period: month prior to the assessment. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Week 6
Population: ITT; N = Subjects who were randomized and received at least one dose of study drug; baseline n = subjects who were randomized and received at least one dose of study drug, had baseline and post-baseline values.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
scores on scale
  Physical Functioning | 3.6 (3.50) | 0.5 (3.71) | 2.4 (3.42) | -0.4 (3.93) | 2.9 (3.52) | 3.6 (3.62)
  Role-Physical | 1.1 (4.24) | 7.0 (4.49) | 7.5 (4.14) | 7.7 (4.77) | 0.9 (4.24) | 9.6 (4.40)
  Bodily Pain | 6.9 (4.16) | 15.8 (4.41) | 12.9 (4.07) | 16.9 (4.87) | 13.3 (4.17) | 18.1 (4.31)
  General Health | 6.5 (2.81) | 5.2 (3.05) | 4.0 (2.75) | 7.5 (3.15) | 3.6 (2.82) | 5.9 (2.90)
  Vitality | 7.4 (3.98) | 11.1 (4.18) | 9.9 (3.86) | 18.5 (4.46) | 11.7 (3.95) | 13.9 (4.08)
  Social Functioning | 7.8 (3.98) | 8.3 (4.20) | 4.8 (3.88) | 4.4 (4.47) | 9.5 (4.00) | 15.6 (4.10)
  Role-Emotional | -2.1 (4.16) | 6.7 (4.38) | 7.8 (4.05) | 1.0 (4.63) | 8.1 (4.13) | 12.7 (4.31)
  Mental Health | 2.9 (3.49) | 1.0 (3.68) | 3.6 (3.43) | 7.6 (3.90) | 3.7 (3.47) | 10.7 (3.59)
  Summary Physical Score | 4.5 (2.83) | 7.4 (3.02) | 6.7 (2.77) | 8.2 (3.29) | 5.6 (2.85) | 9.7 (2.94)
  Summary Emotional Score | 3.7 (3.33) | 6.9 (3.51) | 6.7 (3.24) | 8.2 (3.72) | 8.5 (3.32) | 13.5 (3.43)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; Physical Functioning: Least Squares mean difference. LS Mean, Std. Error, 95% CI and P-value are from an analysis of covariance (ANCOVA) with treatment and geographic region as main effects and baseline value as covariate in the model; Test type: Superiority or Other; p = 0.5384, ANCOVA; Mean Difference (Final Values) = -3.1, 95% CI [-13.2 to 7.0]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.8015, ANCOVA; Mean Difference (Final Values) = -1.2, 95% CI [-10.9 to 8.5]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.4429, ANCOVA; Mean Difference (Final Values) = -4.1, 95% CI [-14.5 to 6.4]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.8860, ANCOVA; Mean Difference (Final Values) = -0.7, 95% CI [-10.5 to 9.1]
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.9963, ANCOVA; Mean Difference (Final Values) = -0.0, 95% CI [-10.0 to 9.9]
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 50 mg; Role-Physical: Least Squares mean difference. LS Mean, Std. Error, 95% CI and P-value are from an analysis of covariance (ANCOVA) with treatment and geographic region as main effects and baseline value as covariate in the model; Test type: Superiority or Other; p = 0.3421, ANCOVA; Mean Difference (Final Values) = 5.9, 95% CI [-6.3 to 18.1]
Statistical Analysis 7: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 19, analysis 6]; Test type: Superiority or Other; p = 0.2849, ANCOVA; Mean Difference (Final Values) = 6.4, 95% CI [-5.4 to 18.1]
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 19, analysis 6]; Test type: Superiority or Other; p = 0.3058, ANCOVA; Mean Difference (Final Values) = 6.6, 95% CI [-6.1 to 19.2]
Statistical Analysis 9: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 19, analysis 6]; Test type: Superiority or Other; p = 0.9604, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI [-12.1 to 11.5]
Statistical Analysis 10: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 19, analysis 6]; Test type: Superiority or Other; p = 0.1661, ANCOVA; Mean Difference (Final Values) = 8.5, 95% CI [-3.6 to 20.6]
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 50 mg; Bodily Pain: Least Squares mean difference. LS Mean, Std. Error, 95% CI and P-value are from an analysis of covariance (ANCOVA) with treatment and geographic region as main effects and baseline value as covariate in the model; Test type: Superiority or Other; p = 0.1441, ANCOVA; Mean Difference (Final Values) = 8.9, 95% CI [-3.1 to 20.9]
Statistical Analysis 12: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 19, analysis 11]; Test type: Superiority or Other; p = 0.3076, ANCOVA; Mean Difference (Final Values) = 6.0, 95% CI [-5.6 to 17.5]
Statistical Analysis 13: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 19, analysis 11]; Test type: Superiority or Other; p = 0.1209, ANCOVA; Mean Difference (Final Values) = 10.0, 95% CI [-2.7 to 22.7]
Statistical Analysis 14: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 19, analysis 11]; Test type: Superiority or Other; p = 0.2791, ANCOVA; Mean Difference (Final Values) = 6.4, 95% CI [-5.3 to 18.0]
Statistical Analysis 15: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 19, analysis 11]; Test type: Superiority or Other; p = 0.0644, ANCOVA; Mean Difference (Final Values) = 11.2, 95% CI [-0.7 to 23.0]
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 50 mg; General Health: Least Squares mean difference. LS Mean, Std. Error, 95% CI and P-value are from an analysis of covariance (ANCOVA) with treatment and geographic region as main effects and baseline value as covariate in the model; Test type: Superiority or Other; p = 0.7544, ANCOVA; Mean Difference (Final Values) = -1.3, 95% CI [-9.5 to 6.9]
Statistical Analysis 17: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 19, analysis 16]; Test type: Superiority or Other; p = 0.5142, ANCOVA; Mean Difference (Final Values) = -2.6, 95% CI [-10.3 to 5.2]
Statistical Analysis 18: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 19, analysis 16]; Test type: Superiority or Other; p = 0.8158, ANCOVA; Mean Difference (Final Values) = 1.0, 95% CI [-7.4 to 9.4]
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 19, analysis 16]; Test type: Superiority or Other; p = 0.4599, ANCOVA; Mean Difference (Final Values) = -2.9, 95% CI [-10.8 to 4.9]
Statistical Analysis 20: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 19, analysis 16]; Test type: Superiority or Other; p = 0.8636, ANCOVA; Mean Difference (Final Values) = -0.7, 95% CI [-8.7 to 7.3]
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 50 mg; Vitality: Least Squares mean difference. LS Mean, Std. Error, 95% CI and P-value are from an analysis of covariance (ANCOVA) with treatment and geographic region as main effects and baseline value as covariate in the model; Test type: Superiority or Other; p = 0.5281, ANCOVA; Mean Difference (Final Values) = 3.7, 95% CI [-7.8 to 15.1]
Statistical Analysis 22: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 19, analysis 21]; Test type: Superiority or Other; p = 0.6566, ANCOVA; Mean Difference (Final Values) = 2.5, 95% CI [-8.5 to 13.5]
Statistical Analysis 23: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 19, analysis 21]; Test type: Superiority or Other; p = 0.0677, ANCOVA; Mean Difference (Final Values) = 11.1, 95% CI [-0.8 to 23.0]
Statistical Analysis 24: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 19, analysis 21]; Test type: Superiority or Other; p = 0.4443, ANCOVA; Mean Difference (Final Values) = 4.3, 95% CI [-6.8 to 15.4]
Statistical Analysis 25: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 19, analysis 21]; Test type: Superiority or Other; p = 0.2543, ANCOVA; Mean Difference (Final Values) = 6.5, 95% CI [-4.7 to 17.7]
Statistical Analysis 26: Comparison: Placebo vs Pregabalin 50 mg; Social Functioning: Least Squares mean difference. LS Mean, Std. Error, 95% CI and P-value are from an analysis of covariance (ANCOVA) with treatment and geographic region as main effects and baseline value as covariate in the model; Test type: Superiority or Other; p = 0.9416, ANCOVA; Mean Difference (Final Values) = 0.4, 95% CI [-11.0 to 11.9]
Statistical Analysis 27: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 19, analysis 26]; Test type: Superiority or Other; p = 0.5824, ANCOVA; Mean Difference (Final Values) = -3.1, 95% CI [-14.1 to 7.9]
Statistical Analysis 28: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 19, analysis 26]; Test type: Superiority or Other; p = 0.5668, ANCOVA; Mean Difference (Final Values) = -3.4, 95% CI [-15.3 to 8.4]
Statistical Analysis 29: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 19, analysis 26]; Test type: Superiority or Other; p = 0.7769, ANCOVA; Mean Difference (Final Values) = 1.6, 95% CI [-9.6 to 12.8]
Statistical Analysis 30: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 19, analysis 26]; Test type: Superiority or Other; p = 0.1753, ANCOVA; Mean Difference (Final Values) = 7.8, 95% CI [-3.5 to 19.1]
Statistical Analysis 31: Comparison: Placebo vs Pregabalin 50 mg; Role-Emotional: Least Squares mean difference. LS Mean, Std. Error, 95% CI and P-value are from an analysis of covariance (ANCOVA) with treatment and geographic region as main effects and baseline value as covariate in the model; Test type: Superiority or Other; p = 0.1508, ANCOVA; Mean Difference (Final Values) = 8.7, 95% CI [-3.2 to 20.7]
Statistical Analysis 32: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 19, analysis 31]; Test type: Superiority or Other; p = 0.0916, ANCOVA; Mean Difference (Final Values) = 9.9, 95% CI [-1.6 to 21.4]
Statistical Analysis 33: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 19, analysis 31]; Test type: Superiority or Other; p = 0.6222, ANCOVA; Mean Difference (Final Values) = 3.1, 95% CI [-9.2 to 15.4]
Statistical Analysis 34: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 19, analysis 31]; Test type: Superiority or Other; p = 0.0850, ANCOVA; Mean Difference (Final Values) = 10.2, 95% CI [-1.4 to 21.8]
Statistical Analysis 35: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 19, analysis 31]; Test type: Superiority or Other; p = 0.0154, ANCOVA; Mean Difference (Final Values) = 14.8, 95% CI [2.9 to 26.7]
Statistical Analysis 36: Comparison: Placebo vs Pregabalin 50 mg; Mental Health: Least Squares mean difference. LS Mean, Std. Error, 95% CI and P-value are from an analysis of covariance (ANCOVA) with treatment and geographic region as main effects and baseline value as covariate in the model; Test type: Superiority or Other; p = 0.7201, ANCOVA; Mean Difference (Final Values) = -1.8, 95% CI [-11.9 to 8.2]
Statistical Analysis 37: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 19, analysis 36]; Test type: Superiority or Other; p = 0.8875, ANCOVA; Mean Difference (Final Values) = 0.7, 95% CI [-9.1 to 10.5]
Statistical Analysis 38: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 19, analysis 36]; Test type: Superiority or Other; p = 0.3735, ANCOVA; Mean Difference (Final Values) = 4.7, 95% CI [-5.7 to 15.1]
Statistical Analysis 39: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 19, analysis 36]; Test type: Superiority or Other; p = 0.8621, ANCOVA; Mean Difference (Final Values) = 0.9, 95% CI [-8.9 to 10.6]
Statistical Analysis 40: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 19, analysis 36]; Test type: Superiority or Other; p = 0.1203, ANCOVA; Mean Difference (Final Values) = 7.9, 95% CI [-2.1 to 17.8]
Statistical Analysis 41: Comparison: Placebo vs Pregabalin 50 mg; Summary Physical Score: Least Squares mean difference. LS Mean, Std. Error, 95% CI and P-value are from an analysis of covariance (ANCOVA) with treatment and geographic region as main effects and baseline value as covariate in the model; Test type: Superiority or Other; p = 0.4966, ANCOVA; Mean Difference (Final Values) = 2.8, 95% CI [-5.4 to 11.0]
Statistical Analysis 42: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 19, analysis 41]; Test type: Superiority or Other; p = 0.5776, ANCOVA; Mean Difference (Final Values) = 2.2, 95% CI [-5.6 to 10.1]
Statistical Analysis 43: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 19, analysis 41]; Test type: Superiority or Other; p = 0.3955, ANCOVA; Mean Difference (Final Values) = 3.7, 95% CI [-4.9 to 12.3]
Statistical Analysis 44: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 19, analysis 41]; Test type: Superiority or Other; p = 0.7994, ANCOVA; Mean Difference (Final Values) = 1.0, 95% CI [-6.9 to 9.0]
Statistical Analysis 45: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 19, analysis 41]; Test type: Superiority or Other; p = 0.2073, ANCOVA; Mean Difference (Final Values) = 5.2, 95% CI [-2.9 to 13.2]
Statistical Analysis 46: Comparison: Placebo vs Pregabalin 50 mg; Summary Emotional Score: Least Squares mean difference. LS Mean, Std. Error, 95% CI and P-value are from an analysis of covariance (ANCOVA) with treatment and geographic region as main effects and baseline value as covariate in the model; Test type: Superiority or Other; p = 0.5148, ANCOVA; Mean Difference (Final Values) = 3.2, 95% CI [-6.4 to 12.8]
Statistical Analysis 47: Comparison: Placebo vs Pregabalin 100 mg; [analysis description as in outcome 19, analysis 46]; Test type: Superiority or Other; p = 0.5255, ANCOVA; Mean Difference (Final Values) = 3.0, 95% CI [-6.3 to 12.2]
Statistical Analysis 48: Comparison: Placebo vs Pregabalin 150 mg; [analysis description as in outcome 19, analysis 46]; Test type: Superiority or Other; p = 0.3793, ANCOVA; Mean Difference (Final Values) = 4.4, 95% CI [-5.5 to 14.4]
Statistical Analysis 49: Comparison: Placebo vs Pregabalin 300 mg; [analysis description as in outcome 19, analysis 46]; Test type: Superiority or Other; p = 0.3120, ANCOVA; Mean Difference (Final Values) = 4.8, 95% CI [-4.5 to 14.1]
Statistical Analysis 50: Comparison: Placebo vs Pregabalin 450 mg; [analysis description as in outcome 19, analysis 46]; Test type: Superiority or Other; p = 0.0442, ANCOVA; Mean Difference (Final Values) = 9.7, 95% CI [0.3 to 19.2]

20. Secondary Outcome: Medical Outcomes Study Short Form 36 (SF-36); Number of Subjects With Self-Evaluated Change in Health Status Scores
Description: Subject-rated measure of health status comprised of 36 items: 8 subscale scores (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health), 2 summary scores (physical component and mental component), and a self-evaluated change in health status. Self-evaluated change in health status: 5 Likert-type response categories ranging from "much worse now" to much better now." Recall period: month prior to the assessment.
Time Frame: Baseline, Week 6
Population: ITT; N = number of subjects in a treatment group.
Measure: Number; unit: participants
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Number analyzed (Participants) | 23 | 22 | 23 | 22 | 24 | 23
participants
  Baseline: Much Worse than 1 Year Ago | 0 | 3 | 1 | 2 | 3 | 2
  Baseline: Somewhat Worse than 1 Year Ago | 4 | 6 | 3 | 4 | 1 | 3
  Baseline: About the Same as 1 Year Ago | 15 | 9 | 15 | 14 | 14 | 12
  Baseline: Somewhat Better than 1 Year Ago | 2 | 1 | 3 | 0 | 5 | 2
  Baseline: Much Better than 1 Year Ago | 1 | 1 | 1 | 0 | 1 | 2
  Week 6: Much Worse than 1 Year Ago | 1 | 0 | 0 | 0 | 2 | 0
  Week 6: Somewhat Worse than 1 Year Ago | 2 | 3 | 2 | 4 | 3 | 1
  Week 6: About the Same as 1 Year Ago | 11 | 12 | 10 | 11 | 12 | 10
  Week 6: Somewhat Better than 1 Year Ago | 4 | 2 | 4 | 1 | 4 | 5
  Week 6: Much Better than 1 Year Ago | 3 | 2 | 6 | 1 | 2 | 4
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 50 mg; CHM test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.4452, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Pregabalin 100 mg; CHM test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.4342, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg; CHM test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.0942, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Pregabalin 300 mg; CHM test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.1873, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Pregabalin 450 mg; CHM test for difference; p-value was adjusted for geographic region at each visit; Test type: Superiority or Other; p = 0.4709, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Arm/Group | Placebo | Pregabalin 50 mg | Pregabalin 100 mg | Pregabalin 150 mg | Pregabalin 300 mg | Pregabalin 450 mg
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/22 | 0/23 | 0/22 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 13/23 | 9/22 | 12/23 | 15/22 | 17/24 | 19/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | Pregabalin 50 mg (N=22) | Pregabalin 100 mg (N=23) | Pregabalin 150 mg (N=22) | Pregabalin 300 mg (N=24) | Pregabalin 450 mg (N=23)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1.45% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | Pregabalin 50 mg (N=22) | Pregabalin 100 mg (N=23) | Pregabalin 150 mg (N=22) | Pregabalin 300 mg (N=24) | Pregabalin 450 mg (N=23)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 4 | 2 | 1 | 2
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0 | 2 | 1
Feeling drunk (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
Feeling jittery (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Feeling of relaxation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
Hangover (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mucosal dryness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Creatinine renal clearance increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Mean cell volume increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 5 | 2 | 7
Dyslalia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 5 | 2 | 2 | 4 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypokinesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1
Post-traumatic headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 6 | 6 | 5
Tunnel vision (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Elevated mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 2 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.